CLINICAL TRIAL: NCT04927065
Title: A Phase 2/3 Study to Evaluate the Immunogenicity and Safety of mRNA Vaccine Boosters for SARS-CoV-2 Variants
Brief Title: A Study to Evaluate the Immunogenicity and Safety of mRNA Vaccine Boosters for SARS-CoV-2 (COVID-19) Variants
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: ModernaTX, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: mRNA-1273-P205
Record Dates: First submitted 2021-06-14; First posted 2021-06-15 (Actual); Results first posted 2025-02-28 (Actual); Last update posted 2025-02-28 (Actual); Status verified 2025-02

CONDITIONS: SARS-CoV-2
Keywords: mRNA-1273; mRNA-1273 vaccine; mRNA-1273.211; mRNA-1273.617.2; mRNA-1273.213; mRNA-1273.529; mRNA-1273.214; mRNA-1273.815; mRNA-1273.231; SARS-CoV-2; SARS-CoV-2 Vaccine; Coronavirus; Virus Diseases; Messenger RNA; COVID 19; COVID 19 Vaccine; Moderna
MeSH Terms: conditions — Coronavirus Infections; Virus Diseases; COVID-19 | interventions — 2019-nCoV Vaccine mRNA-1273; mRNA-1273.214 COVID-19 vaccine

STUDY DESIGN:
Intervention Model Description: Parts A-H: Sequential Part J: Parallel (participants were randomized to receive either mRNA-1273.815 or mRNA-1273.231)
Masking Description: Parts A-H: non-randomized Part J: randomized
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (14):
- Part A.1: mRNA-1273.211 50 μg (Experimental): Participants will receive 1 intramuscular booster dose of 50 micrograms (μg) of mRNA-1273.211 on Day 1.
  Interventions: Biological: mRNA-1273.211
- Part A.1: mRNA-1273.211 100 μg (Experimental): Participants will receive 1 intramuscular booster dose of 100 μg of mRNA-1273.211 on Day 1.
  Interventions: Biological: mRNA-1273.211
- Part B: mRNA-1273 100 μg (Experimental): Participants will receive 1 intramuscular booster dose of 100 μg of mRNA-1273 on Day 1.
  Interventions: Biological: mRNA-1273
- Part C: mRNA-1273.617.2 100 μg (Experimental): Participants will receive 1 intramuscular booster dose of 100 μg of mRNA-1273.617.2 on Day 1.
  Interventions: Biological: mRNA-1273.617.2
- Part C: mRNA-1273.617.2 50 μg (Experimental): Participants will receive 1 intramuscular booster dose of 50 μg of mRNA-1273.617.2 on Day 1.
  Interventions: Biological: mRNA-1273.617.2
- Part D: mRNA-1273.213 50 μg (Experimental): Participants will receive 1 intramuscular booster dose of 50 μg of mRNA-1273.213 on Day 1.
  Interventions: Biological: mRNA-1273.213
- Part D: mRNA-1273.213 100 μg (Experimental): Participants will receive 1 intramuscular booster dose of 100 μg of mRNA-1273.213 on Day 1.
  Interventions: Biological: mRNA-1273.213
- Part E: mRNA-1273.213 100 μg (Experimental): Participants will receive 1 intramuscular booster dose of 100 μg of mRNA-1273.213 on Day 1.
  Interventions: Biological: mRNA-1273.213
- Part F Cohort 1: mRNA-1273.529 50 μg (Experimental): Participants will receive 1 intramuscular first booster dose of 50 μg of mRNA-1273.529 on Day 1.
  Interventions: Biological: mRNA-1273.529
- Part F Cohort 2: mRNA-1273.529 50 μg and mRNA-1273 50 μg (Experimental): Participants will receive 1 intramuscular second booster dose of 50 μg of mRNA-1273.529 or mRNA-1273 enrolled sequentially (after receiving a primary series of mRNA-1273 and a single booster dose of mRNA-1273 50 μg) on Day 1.
  Interventions: Biological: mRNA-1273; Biological: mRNA-1273.529
- Part G: mRNA-1273.214 50 μg (Experimental): Participants will receive 1 intramuscular second booster dose of mRNA-1273.214 50 μg on Day 1.
  Interventions: Biological: mRNA-1273.214
- Part A.2: mRNA-1273.214 50 μg (Experimental): Participants will receive 1 intramuscular booster dose of 50 μg of mRNA-1273.214 on Day 1.
  Interventions: Biological: mRNA-1273.214
- Part H: mRNA-1273.222 50 μg (Experimental): Participants will receive 1 intramuscular second booster dose of 50 μg of mRNA-1273.222 on Day 1.
  Interventions: Biological: mRNA-1273.222
- Part J: mRNA-1273.815 or mRNA-1273.231 (Experimental): Participants will receive 1 intramuscular booster dose of 50 μg of mRNA-1273.815 or 50 ug of mRNA-1273.231 on Day 1.
  Interventions: Biological: mRNA-1273.815; Biological: mRNA-1273.231

INTERVENTIONS:
Biological: mRNA-1273.211 — Sterile liquid for injection
  Arms: Part A.1: mRNA-1273.211 100 μg; Part A.1: mRNA-1273.211 50 μg
Biological: mRNA-1273 — Sterile liquid for injection
  Arms: Part B: mRNA-1273 100 μg; Part F Cohort 2: mRNA-1273.529 50 μg and mRNA-1273 50 μg
Biological: mRNA-1273.617.2 — Sterile liquid for injection
  Arms: Part C: mRNA-1273.617.2 100 μg; Part C: mRNA-1273.617.2 50 μg
Biological: mRNA-1273.213 — Sterile liquid for injection
  Arms: Part D: mRNA-1273.213 100 μg; Part D: mRNA-1273.213 50 μg; Part E: mRNA-1273.213 100 μg
Biological: mRNA-1273.529 — Sterile liquid for injection
  Arms: Part F Cohort 1: mRNA-1273.529 50 μg; Part F Cohort 2: mRNA-1273.529 50 μg and mRNA-1273 50 μg
Biological: mRNA-1273.214 — Sterile liquid for injection
  Arms: Part A.2: mRNA-1273.214 50 μg; Part G: mRNA-1273.214 50 μg
Biological: mRNA-1273.222 — Sterile liquid for injection
  Arms: Part H: mRNA-1273.222 50 μg
Biological: mRNA-1273.815 — Sterile liquid for injection
  Arms: Part J: mRNA-1273.815 or mRNA-1273.231
Biological: mRNA-1273.231 — Sterile liquid for injection
  Arms: Part J: mRNA-1273.815 or mRNA-1273.231

SUMMARY:
This is a study to evaluate the immunogenicity, safety, and reactogenicity of mRNA-1273.211, mRNA-1273, mRNA-1273.617.2, mRNA-1273.213, mRNA-1273.529, mRNA-1273.214, mRNA-1273.222, mRNA-1273.815, and mRNA-1273.231 administered as booster doses.

DETAILED DESCRIPTION:
This clinical study will consist of 9 parts: A (1 and 2), B, C, D, E, F, G, H, and J.

Part A.1 will evaluate 2 dose levels of the mRNA-1273.211 vaccine when administered as a single booster dose to adult participants of the mRNA-1273-P301 (COVE [NCT04470427]) study who have previously received 2 doses of mRNA-1273.

Part A.2 will evaluate the immunogenicity, safety, and reactogenicity of the mRNA-1273.214 vaccine candidate when administered as a second booster dose to adult participants of the mRNA-1273-P205 study who have previously received 2 doses of mRNA-1273 as a primary series and a first booster of (50 μg total mRNA content) of the mRNA-1273.211 in Part A.1 of this study.

Part B will evaluate the mRNA-1273 vaccine when administered as a single booster dose to adult participants of the mRNA-1273-P301 (COVE [NCT04470427]) study who have previously received 2 doses of mRNA-1273.

Part C will evaluate 2 dose levels of the mRNA-1273.617.2 vaccine when administered as a single booster dose to adult participants of the mRNA-1273-P301 (COVE [NCT04470427]) study who have previously received 2 doses of mRNA-1273.

Part D will evaluate 2 dose levels of the mRNA-1273.213 vaccine when administered as a single booster dose to adult participants of the mRNA-1273-P301 (COVE [NCT04470427]) study who have previously received 2 doses of mRNA-1273.

Part E will be enrolled at a single clinical study site. Part E will evaluate the mRNA-1273.213 vaccine when administered as a single booster dose to adult participants who have previously received 2 doses of any SARS-CoV-2 mRNA authorized vaccine, including mRNA-1273.

Part F will consist of 2 cohorts: Cohort 1 will consist of adults who have previously received 2 doses of mRNA-1273 as primary series. Cohort 1 will evaluate the mRNA-1273.529 vaccine as a single booster dose. Cohort 2 will consist of adults who have previously received 2 doses of mRNA-1273 as a primary series and a single booster dose of mRNA-1273 in study mRNA-1273-P301 (COVE [NCT04470427]) or under the emergency use authorization (EUA). Cohort 2 will evaluate the mRNA-1273.529 and mRNA-1273 vaccines as a single booster dose.

Part G will evaluate the mRNA1273.214 vaccine candidate when administered as a second booster dose to adults who have previously received 2 doses of mRNA-1273 as a primary series and a single booster dose of mRNA-1273.

Part H will evaluate the immunogenicity, safety, and reactogenicity of the mRNA- 1273.222 vaccine candidate when administered as a second booster dose to adults who have previously received 2 doses of mRNA-1273 as a primary series and a single booster dose of mRNA-1273.

Part J will evaluate mRNA-1273.815 and mRNA-1273.231 when administered as a booster dose to adults who previously received a primary series of mRNA vaccine, a first booster dose of a monovalent mRNA vaccine, and a second booster dose of a bivalent mRNA vaccine against SARS-COV-2.

ELIGIBILITY:
Key Inclusion Criteria:

* For female participants of childbearing potential: negative pregnancy test, adequate contraception or has abstained from all activities that could result in pregnancy for at least 28 days prior to Day 1, agreement to continue adequate contraception or abstinence through 3 months following the vaccination, and not currently breastfeeding.
* Participants must have been either previously enrolled in the mRNA-1273-P301 (COVE) study, must have received 2 doses of mRNA-1273 in that study, with their second dose at least 6 months prior to enrollment in this study (mRNA-1273-P205), and must be currently enrolled and compliant in that study (that is, has not withdrawn or discontinued early); or participant must have received 2 doses of mRNA-1273 under the EUA with their second dose at least 6 months prior to enrollment in mRNA-1273-P205; or have received a 2 dose primary series of mRNA-1273 followed by a 50 μg booster dose of mRNA-1273 in the mRNA-1273-P301 (COVE) study or under EUA at least 3 months prior to enrolment in mRNA-1273-P205; and able to provide proof of vaccination status at the time of screening (Day 1); or for enrollment in Part A.2, participant must be currently enrolled and compliant in Part A.1 of the mRNA 1273 P205 study and must have received their first booster dose of mRNA 1273.211 50 μg; or for enrollment in Part J, participant must meet at least 1 of the following criteria: completed enrollment in Part H of the mRNA-1273-P205 study; or received a 2-dose primary series of mRNA-1273 (100 μg) followed by a 50 μg booster dose of mRNA-1273 in the mRNA-1273-P301 (COVE) study or under EUA, followed by a 50 μg booster dose of mRNA-1273.222 under EUA at least 3 months prior to enrollment in Part J of mRNA-1273-P205; or previously received a 2-dose primary series of mRNA vaccine against SARS-CoV-2 followed by a booster dose of a monovalent mRNA vaccine, followed by a second booster dose of a bivalent mRNA vaccine. Participants in Part J must also provide proof of vaccination status at the time of screening (Day 0 or Day 1).

Key Exclusion Criteria:

* Significant exposure to someone with SARS-CoV-2 infection or COVID-19 in the past 14 days, as defined by the US Centers for Disease Control and Prevention (CDC) as a close contact of someone who has had COVID-19.
* Known history of SARS-CoV-2 infection within 3 months prior to enrollment.
* Is acutely ill or febrile (temperature ≥38.0°Celsius/[100.4°Fahrenheit]) less than 72 hours prior to or at the Screening Visit (Day 0) or Day 1.
* Has a medical, psychiatric, or occupational condition that may pose additional risk as a result of participation, or that could interfere with safety assessments or interpretation of results according to the investigator's judgment.
* Has received systemic immunosuppressants or immune-modifying drugs for >14 days in total within 6 months prior to Screening (for corticosteroids ≥10 milligrams (mg)/day of prednisone equivalent) or is anticipating the need for immunosuppressive treatment at any time during participation in the study.
* Known or suspected allergy or history of anaphylaxis, urticaria, or other significant AR to the vaccine or its excipients.
* Has a documented history of myocarditis or pericarditis within 2 months prior to Screening Visit (Day 0).
* Has received or plans to receive any licensed vaccine ≤28 days prior to the injection (Day 1) or a licensed vaccine within 28 days before or after they study injection, with the exception of influenza vaccines, which may be given 14 days before or after receipt of a study vaccine.
* Has received systemic immunoglobulins or blood products within 3 months prior to the Screening Visit (Day 0) or plans for receipt during the study.
* Has donated ≥450 milliliters (mL) of blood products within 28 days prior to the Screening Visit (Day 0) or plans to donate blood products during the study.
* Is currently experiencing an SAE in Study mRNA-1273-P301 (COVE) at the time of screening for this study.

Note: Other inclusion and exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5161 (Actual)
Dates: Start 2021-05-28 (Actual); Primary Completion 2023-11-17 (Actual); Study Completion 2023-11-17 (Actual)

CONTACTS AND LOCATIONS:
Locations (23):
- United States (23):
  - Benchmark Research (California), Sacramento, California
  - Research Centers of America, Hollywood, Florida
  - Jacksonville Center For Clinical Research, Jacksonville, Florida
  - Meridian Clinical Research-(Savannah Georgia), Savannah, Georgia
  - Meridian Clinical Research (Iowa), Sioux City, Iowa
  - Johnson County Clinical Trials, Lenexa, Kansas
  - Meridian Clinical Research-(Baton Rouge, Louisiana), Baton Rouge, Louisiana
  - Benchmark Research, Metairie, Louisiana
  - Meridian Clinical Research-(Rockville Maryland), Rockville, Maryland
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Washington State University, St Louis, Missouri
  - Sundance Clinical Research, St Louis, Missouri
  - Meridian Clinical Research (Grand Island, Nebraska), Grand Island, Nebraska
  - Meridian Clinical Research (Norfolk-Nebraska), Norfolk, Nebraska
  - Meridian Clinical Research-(Omaha Nebraska), Omaha, Nebraska
  - Meridian Clinical Research, LLC, New York, New York
  - Trial Management Associates, Wilmington, North Carolina
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Benchmark Research - Austin - HyperCore, Austin, Texas
  - Tekton Research, Inc., Austin, Texas
  - Benchmark Research - Fort Worth - HyperCore, Fort Worth, Texas
  - Texas Center for Drug Development, Inc., Houston, Texas
  - DM Clinical Research, Tomball, Texas

REFERENCES:
- [Derived] Chalkias S, Whatley JL, Eder F, Essink B, Khetan S, Bradley P, Brosz A, McGhee N, Tomassini JE, Chen X, Zhao X, Sutherland A, Shen X, Girard B, Edwards DK, Feng J, Zhou H, Walsh S, Montefiori DC, Baden LR, Miller JM, Das R. Original SARS-CoV-2 monovalent and Omicron BA.4/BA.5 bivalent COVID-19 mRNA vaccines: phase 2/3 trial interim results. Nat Med. 2023 Sep;29(9):2325-2333. doi: 10.1038/s41591-023-02517-y. Epub 2023 Aug 31. PMID 37653342
- [Derived] Chalkias S, Harper C, Vrbicky K, Walsh SR, Essink B, Brosz A, McGhee N, Tomassini JE, Chen X, Chang Y, Sutherland A, Montefiori DC, Girard B, Edwards DK, Feng J, Zhou H, Baden LR, Miller JM, Das R. A Bivalent Omicron-Containing Booster Vaccine against Covid-19. N Engl J Med. 2022 Oct 6;387(14):1279-1291. doi: 10.1056/NEJMoa2208343. Epub 2022 Sep 16. PMID 36112399
- [Derived] Chalkias S, Schwartz H, Nestorova B, Feng J, Chang Y, Zhou H, Dutko FJ, Edwards DK, Montefiori D, Pajon R, Leav B, Miller JM, Das R. Safety and Immunogenicity of a 100 mug mRNA-1273 Vaccine Booster for Severe Acute Respiratory Syndrome Coronavirus-2 (SARS-CoV-2). medRxiv [Preprint]. 2022 Mar 7:2022.03.04.22271830. doi: 10.1101/2022.03.04.22271830. PMID 35291289

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 135 participants from Part A.1 rolled over to Part A.2. 87 participants from Part H rolled over to Part J. Therefore, a total number of enrolled and treated participants in the study = 5161.
Groups:
- Part A.1: mRNA-1273.211 50 μg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (NCT04470427; COVE), received a single intramuscular (IM) booster dose of 50 micrograms (μg) of mRNA-1273.211 on Day 1 of Part A.1.
- Part A.1: mRNA-1273.211 100 μg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (COVE), received a single IM booster dose of 100 μg of mRNA-1273.211 on Day 1 of Part A.1.
- Part A.2: mRNA-1273.214 50 μg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (COVE) and a first booster dose of 50 μg of the mRNA-1273.211 in Part A.1 of this study, received a second IM booster dose of 50 μg of mRNA-1273.214 on Day 1 of Part A.2.
- Part B: mRNA-1273 100 μg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (COVE), received a single IM booster dose of 100 μg of mRNA-1273 on Day 1 of Part B.
- Part C: mRNA-1273.617.2 50 μg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (COVE) or under the Emergency Use Authorization (EUA), received a single IM booster dose of 50 μg of mRNA-1273.617.2 on Day 1 of Part C.
- Part C: mRNA-1273.617.2 100 μg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (COVE) or under the EUA, received a single IM booster dose of 100 μg of mRNA-1273.617.2 on Day 1 of Part C.
- Part D: mRNA-1273.213 50 μg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (COVE) or under the EUA, received a single IM booster dose of 50 μg of mRNA-1273.213 on Day 1 of Part D.
- Part D: mRNA-1273.213 100 μg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (COVE) or under the EUA, received a single IM booster dose of 100 μg of mRNA-1273.213 on Day 1 of Part D.
- Part E: mRNA-1273.213 100 μg: Participants who had previously received 2 doses of any SARS-CoV-2 mRNA authorized vaccine as a primary series (with a subset of enrolled participants who previously received Moderna's mRNA-1273 authorized vaccine as a primary series), received a single IM booster dose of 100 μg of mRNA-1273.213 on Day 1 of Part E.
- Part F (Cohort 1): mRNA-1273.529 50 μg: Participants who had previously received 2 doses of mRNA-1273 as a primary series, received a single IM booster dose of 50 μg of mRNA-1273.529 on Day 1 of Part F.
- Part F (Cohort 2): mRNA-1273 50 μg: Participants who had previously received 2 doses of mRNA-1273 100 μg as a primary series and a single booster dose of mRNA-1273 50 μg in Study mRNA-1273-P301 (COVE) or under the EUA, received a second IM booster dose of 50 μg of mRNA-1273 on Day 1 of Part F.
- Part F (Cohort 2): mRNA-1273.529 50 μg: Participants who had previously received 2 doses of mRNA-1273 100 μg as a primary series and a single booster dose of mRNA-1273 50 μg in Study mRNA-1273-P301 (COVE) or under the EUA, received a second IM booster dose of 50 μg of mRNA-1273.529 on Day 1 of Part F.
- Part G: mRNA-1273.214 50 μg: Participants who had previously received 2 doses of mRNA-1273 100 μg as a primary series and a single booster dose of mRNA-1273 50 μg, received a second IM booster dose of mRNA-1273.214 50 μg on Day 1 of Part G.
- Part H: mRNA-1273.222 50 μg: Participants who had previously received 2 doses of mRNA-1273 100 μg as a primary series and a single booster dose of mRNA-1273 50 μg, received a second IM booster dose of 50 μg of mRNA-1273.222 on Day 1 of Part H.
- Part J: mRNA-1273.231 50 μg: Participants who previously received a primary series of mRNA vaccine, a first booster dose of a monovalent mRNA vaccine, and a second booster dose of a bivalent mRNA vaccine against SARS-CoV-2, received a third IM booster dose of 50 μg of mRNA-1273.231 on Day 1 of Part J.
- Part J: mRNA-1273.815 50 μg: Participants who previously received a primary series of mRNA vaccine, a first booster dose of a monovalent mRNA vaccine, and a second booster dose of a bivalent mRNA vaccine against SARS-CoV-2, received a third IM booster dose of 50 ug of mRNA-1273.815 on Day 1 of Part J.
Period: First Booster
Arm/Group | Part A.1: mRNA-1273.211 50 μg | Part A.1: mRNA-1273.211 100 μg | Part A.2: mRNA-1273.214 50 μg | Part B: mRNA-1273 100 μg | Part C: mRNA-1273.617.2 50 μg | Part C: mRNA-1273.617.2 100 μg | Part D: mRNA-1273.213 50 μg | Part D: mRNA-1273.213 100 μg | Part E: mRNA-1273.213 100 μg | Part F (Cohort 1): mRNA-1273.529 50 μg | Part F (Cohort 2): mRNA-1273 50 μg | Part F (Cohort 2): mRNA-1273.529 50 μg | Part G: mRNA-1273.214 50 μg | Part H: mRNA-1273.222 50 μg | Part J: mRNA-1273.231 50 μg | Part J: mRNA-1273.815 50 μg
Started (Full Analysis Set) | 300 | 593 | 0 | 305 | 581 | 586 | 327 | 583 | 42 | 133 | 0 | 0 | 0 | 0 | 0 | 0
Safety Set (All participants who received investigational product (IP).) | 300 | 593 | 0 | 305 | 581 | 586 | 327 | 583 | 42 | 133 | 0 | 0 | 0 | 0 | 0 | 0
Solicited Safety Set (All participants who received IP and contributed any solicited adverse reaction (AR) data.) | 298 | 591 | 0 | 303 | 577 | 583 | 327 | 583 | 42 | 133 | 0 | 0 | 0 | 0 | 0 | 0
Per-Protocol Immunogenicity SARS-CoV-2 Negative Set (PPIS-Neg) (All participants who received the planned dose of study injection per schedule; had pre-booster and Day 29 nAb data (for Parts A.1, A.2, B, C, D, F, G, and H); had pre-booster and Day 15 nAb data (for Part J); had no major protocol deviations that impacted key or critical data; had no previous HIV infection; and who had no serologic or virologic evidence of SARS-CoV-2 infection at baseline.) | 295 | 563 | 0 | 245 | 489 | 547 | 250 | 509 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Per-Protocol Immunogenicity Set (PPIS) (All participants who received study injection; had pre-booster and Day 15 nAb data; and who had no major protocol deviations that impacted key or critical data.) | 299 | 576 | 0 | 257 | 537 | 569 | 314 | 543 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 276 | 545 | 0 | 267 | 515 | 536 | 291 | 524 | 38 | 110 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 24 | 48 | 0 | 38 | 66 | 50 | 36 | 59 | 4 | 23 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Death | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 8 | 20 | 0 | 11 | 43 | 30 | 28 | 23 | 4 | 15 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 0 | 3 | 1 | 1 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 4 | 4 | 0 | 3 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 8 | 23 | 0 | 19 | 20 | 15 | 6 | 24 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Other Than Specified | 1 | 1 | 0 | 1 | 2 | 3 | 2 | 6 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0
Period: Second Booster
Arm/Group | Part A.1: mRNA-1273.211 50 μg | Part A.1: mRNA-1273.211 100 μg | Part A.2: mRNA-1273.214 50 μg | Part B: mRNA-1273 100 μg | Part C: mRNA-1273.617.2 50 μg | Part C: mRNA-1273.617.2 100 μg | Part D: mRNA-1273.213 50 μg | Part D: mRNA-1273.213 100 μg | Part E: mRNA-1273.213 100 μg | Part F (Cohort 1): mRNA-1273.529 50 μg | Part F (Cohort 2): mRNA-1273 50 μg | Part F (Cohort 2): mRNA-1273.529 50 μg | Part G: mRNA-1273.214 50 μg | Part H: mRNA-1273.222 50 μg | Part J: mRNA-1273.231 50 μg | Part J: mRNA-1273.815 50 μg
Started (Full Analysis Set) | 0 | 0 | 135 (Participants from Part A.1) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 376 | 375 | 437 | 510 | 0 | 0
Safety Set (All participants who received IP.) | 0 | 0 | 135 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 376 | 375 | 437 | 510 | 0 | 0
Solicited Safety Set (All participants who received IP and contributed any solicited AR data.) | 0 | 0 | 128 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 350 | 372 | 437 | 507 | 0 | 0
PPIS-Neg (All participants who received the planned dose of study injection per schedule; had pre-booster and Day 29 nAb data (for Parts A.1, A.2, B, C, D, F, G, and H); had pre-booster and Day 15 nAb data (for Part J); had no major protocol deviations that impacted key or critical data; had no previous HIV infection; and who had no serologic or virologic evidence of SARS-CoV-2 infection at baseline.) | 0 | 0 | 76 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 258 | 273 | 334 | 209 | 0 | 0
PPIS (All participants who received study injection; had pre-booster and Day 15 nAb data; and who had no major protocol deviations that impacted key or critical data.) | 0 | 0 | 126 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 362 | 358 | 428 | 494 | 0 | 0
Completed | 0 | 0 | 128 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 356 | 345 | 405 | 482 | 0 | 0
Not Completed | 0 | 0 | 7 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 20 | 30 | 32 | 28 | 0 | 0
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 2 | 2 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 14 | 10 | 13 | 16 | 0 | 0
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 1 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 16 | 13 | 9 | 0 | 0
Not completed — Other Than Specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 4 | 0 | 0 | 0
Period: Third Booster
Arm/Group | Part A.1: mRNA-1273.211 50 μg | Part A.1: mRNA-1273.211 100 μg | Part A.2: mRNA-1273.214 50 μg | Part B: mRNA-1273 100 μg | Part C: mRNA-1273.617.2 50 μg | Part C: mRNA-1273.617.2 100 μg | Part D: mRNA-1273.213 50 μg | Part D: mRNA-1273.213 100 μg | Part E: mRNA-1273.213 100 μg | Part F (Cohort 1): mRNA-1273.529 50 μg | Part F (Cohort 2): mRNA-1273 50 μg | Part F (Cohort 2): mRNA-1273.529 50 μg | Part G: mRNA-1273.214 50 μg | Part H: mRNA-1273.222 50 μg | Part J: mRNA-1273.231 50 μg | Part J: mRNA-1273.815 50 μg
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 50 (45 participants rolled over from Part H.) | 50 (42 participants rolled over from Part H.)
Safety Set (All participants who received IP.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 50 | 50
Solicited Safety Set (All participants who received IP and contributed any solicited AR data.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 50 | 50
PPIS-Neg (All participants who received the planned dose of study injection per schedule; had pre-booster and Day 29 nAb data (for Parts A.1, A.2, B, C, D, F, G, and H); had pre-booster and Day 15 nAb data (for Part J); had no major protocol deviations that impacted key or critical data; had no previous HIV infection; and who had no serologic or virologic evidence of SARS-CoV-2 infection at baseline.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 11 | 16
PPIS (All participants who received study injection; had pre-booster and Day 15 nAb data; and who had no major protocol deviations that impacted key or critical data.) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 49 | 49
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 50 | 48
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Set included all participants who received IP. Total number of enrolled and treated participants in the study = 5161. All participants of Part A.2 rolled over from Part A.1 and some participants of Parts J rolled over from Part H. Hence, the baseline characteristics data of Part A.2 and Parts J are reported in a separate row.
Groups:
- Part A.1: mRNA-1273.211 50 μg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (COVE), received a single intramuscular (IM) booster dose of 50 micrograms (μg) of mRNA-1273.211 on Day 1 of Part A.1.
- Part C: mRNA-1273.617.2 50 μg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (COVE) or under the EUA, received a single IM booster dose of 50 μg of mRNA-1273.617.2 on Day 1 of Part C.
- Total: Total of all reporting groups
Arm/Group | Part A.1: mRNA-1273.211 50 μg | Part A.1: mRNA-1273.211 100 μg | Part A.2: mRNA-1273.214 50 μg | Part B: mRNA-1273 100 μg | Part C: mRNA-1273.617.2 50 μg | Part C: mRNA-1273.617.2 100 μg | Part D: mRNA-1273.213 50 μg | Part D: mRNA-1273.213 100 μg | Part E: mRNA-1273.213 100 μg | Part F (Cohort 1): mRNA-1273.529 50 μg | Part F (Cohort 2): mRNA-1273 50 μg | Part F (Cohort 2): mRNA-1273.529 50 μg | Part G: mRNA-1273.214 50 μg | Part H: mRNA-1273.222 50 μg | Part J: mRNA-1273.231 50 μg | Part J: mRNA-1273.815 50 μg | Total
Number analyzed (Participants) | 300 | 593 | 135 | 305 | 581 | 586 | 327 | 583 | 42 | 133 | 376 | 375 | 437 | 510 | 50 | 50 | 5383
Age, Categorical [Count of Participants; unit: Participants] — Population: Baseline characteristics data of Part A.2 and Parts J are reported in a separate row to avoid double-counting of the participants.
  Participants
    All Parts Excluding Part A.2 and Parts J: number analyzed (Participants) | 300 | 593 | 0 | 305 | 581 | 586 | 327 | 583 | 42 | 133 | 376 | 375 | 437 | 510 | 0 | 0 | 5148
    All Parts Excluding Part A.2 and Parts J: <=18 years | 0 | 0 |  | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 |  |  | 0
    All Parts Excluding Part A.2 and Parts J: Between 18 and 65 years | 238 | 447 |  | 216 | 466 | 467 | 292 | 426 | 41 | 115 | 226 | 254 | 263 | 405 |  |  | 3856
    All Parts Excluding Part A.2 and Parts J: >=65 years | 62 | 146 |  | 89 | 115 | 119 | 35 | 157 | 1 | 18 | 150 | 121 | 174 | 105 |  |  | 1292
    Part A.2 and Parts J: number analyzed (Participants) | 0 | 0 | 135 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 50 | 50 | 235
    Part A.2 and Parts J: <=18 years |  |  | 0 |  |  |  |  |  |  |  |  |  |  |  | 0 | 0 | 0
    Part A.2 and Parts J: Between 18 and 65 years |  |  | 112 |  |  |  |  |  |  |  |  |  |  |  | 43 | 39 | 194
    Part A.2 and Parts J: >=65 years |  |  | 23 |  |  |  |  |  |  |  |  |  |  |  | 7 | 11 | 41
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Baseline characteristics data of Part A.2 and Parts J are reported in a separate row to avoid double-counting of the participants.
  Participants
    All Parts Excluding Part A.2 and Parts J: number analyzed (Participants) | 300 | 593 | 0 | 305 | 581 | 586 | 327 | 583 | 42 | 133 | 376 | 375 | 437 | 510 | 0 | 0 | 5148
    All Parts Excluding Part A.2 and Parts J: Female | 167 | 330 |  | 131 | 313 | 287 | 204 | 284 | 23 | 70 | 190 | 173 | 258 | 316 |  |  | 2746
    All Parts Excluding Part A.2 and Parts J: Male | 133 | 263 |  | 174 | 268 | 299 | 123 | 299 | 19 | 63 | 186 | 202 | 179 | 194 |  |  | 2402
    Part A.2 and Parts J: number analyzed (Participants) | 0 | 0 | 135 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 50 | 50 | 235
    Part A.2 and Parts J: Female |  |  | 75 |  |  |  |  |  |  |  |  |  |  |  | 31 | 30 | 136
    Part A.2 and Parts J: Male |  |  | 60 |  |  |  |  |  |  |  |  |  |  |  | 19 | 20 | 99
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics data of Part A.2 and Parts J are reported in a separate row to avoid double-counting of the participants.
  Participants
    All Parts Excluding Part A.2 and Parts J: number analyzed (Participants) | 300 | 593 | 0 | 305 | 581 | 586 | 327 | 583 | 42 | 133 | 376 | 375 | 437 | 510 | 0 | 0 | 5148
    All Parts Excluding Part A.2 and Parts J: Hispanic or Latino | 38 | 51 |  | 66 | 100 | 106 | 32 | 68 | 1 | 17 | 37 | 47 | 46 | 58 |  |  | 667
    All Parts Excluding Part A.2 and Parts J: Not Hispanic or Latino | 262 | 538 |  | 237 | 475 | 474 | 294 | 512 | 41 | 113 | 339 | 324 | 390 | 447 |  |  | 4446
    All Parts Excluding Part A.2 and Parts J: Unknown or Not Reported | 0 | 4 |  | 2 | 6 | 6 | 1 | 3 | 0 | 3 | 0 | 4 | 1 | 5 |  |  | 35
    Part A.2 and Parts J: number analyzed (Participants) | 0 | 0 | 135 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 50 | 50 | 235
    Part A.2 and Parts J: Hispanic or Latino |  |  | 15 |  |  |  |  |  |  |  |  |  |  |  | 6 | 9 | 30
    Part A.2 and Parts J: Not Hispanic or Latino |  |  | 120 |  |  |  |  |  |  |  |  |  |  |  | 43 | 40 | 203
    Part A.2 and Parts J: Unknown or Not Reported |  |  | 0 |  |  |  |  |  |  |  |  |  |  |  | 1 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Baseline characteristics data of Part A.2 and Parts J are reported in a separate row to avoid double-counting of the participants.
  Participants
    All Parts Excluding Part A.2 and Parts J: number analyzed (Participants) | 300 | 593 | 0 | 305 | 581 | 586 | 327 | 583 | 42 | 133 | 376 | 375 | 437 | 510 | 0 | 0 | 5148
    All Parts Excluding Part A.2 and Parts J: American Indian or Alaska Native | 1 | 5 |  | 0 | 5 | 1 | 2 | 3 | 0 | 0 | 1 | 3 | 0 | 1 |  |  | 22
    All Parts Excluding Part A.2 and Parts J: Asian | 9 | 18 |  | 6 | 23 | 51 | 10 | 26 | 2 | 6 | 16 | 14 | 14 | 11 |  |  | 206
    All Parts Excluding Part A.2 and Parts J: Native Hawaiian or Other Pacific Islander | 0 | 1 |  | 0 | 0 | 2 | 1 | 2 | 0 | 0 | 1 | 2 | 0 | 0 |  |  | 9
    All Parts Excluding Part A.2 and Parts J: Black or African American | 19 | 34 |  | 17 | 54 | 32 | 23 | 49 | 1 | 26 | 28 | 21 | 31 | 56 |  |  | 391
    All Parts Excluding Part A.2 and Parts J: White | 257 | 518 |  | 279 | 473 | 481 | 282 | 478 | 38 | 97 | 322 | 325 | 381 | 425 |  |  | 4356
    All Parts Excluding Part A.2 and Parts J: More than one race | 7 | 7 |  | 1 | 7 | 10 | 6 | 12 | 0 | 1 | 2 | 7 | 7 | 8 |  |  | 75
    All Parts Excluding Part A.2 and Parts J: Unknown or Not Reported | 7 | 10 |  | 2 | 19 | 9 | 3 | 13 | 1 | 3 | 6 | 3 | 4 | 9 |  |  | 89
    Part A.2 and Parts J: number analyzed (Participants) | 0 | 0 | 135 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 50 | 50 | 235
    Part A.2 and Parts J: American Indian or Alaska Native |  |  | 1 |  |  |  |  |  |  |  |  |  |  |  | 0 | 0 | 1
    Part A.2 and Parts J: Asian |  |  | 1 |  |  |  |  |  |  |  |  |  |  |  | 2 | 1 | 4
    Part A.2 and Parts J: Native Hawaiian or Other Pacific Islander |  |  | 0 |  |  |  |  |  |  |  |  |  |  |  | 0 | 0 | 0
    Part A.2 and Parts J: Black or African American |  |  | 10 |  |  |  |  |  |  |  |  |  |  |  | 4 | 4 | 18
    Part A.2 and Parts J: White |  |  | 117 |  |  |  |  |  |  |  |  |  |  |  | 41 | 45 | 203
    Part A.2 and Parts J: More than one race |  |  | 2 |  |  |  |  |  |  |  |  |  |  |  | 2 | 0 | 4
    Part A.2 and Parts J: Unknown or Not Reported |  |  | 4 |  |  |  |  |  |  |  |  |  |  |  | 1 | 0 | 5

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Solicited Local and Systemic ARs
Description: Solicited ARs (local and systemic) were collected in an electronic diary (eDiary). Local ARs included: injection site pain, injection site erythema (redness), injection site swelling/induration (hardness), and axillary (underarm) swelling or tenderness ipsilateral to the side of injection. Systemic ARs included: fever, headache, fatigue, myalgia, arthralgia, nausea/vomiting, and chills. All solicited ARs considered causally related to injection were graded 0-4 (per Toxicity Grading Scale for Healthy Adult and Adolescent Volunteers Enrolled in Preventive Vaccine Clinical Trials); lower score indicates lower severity, and a higher score indicates greater severity. The Investigator reviewed whether the solicited AR was also to be recorded as an adverse event (AE). A Summary of serious AEs (SAEs) and nonserious AEs ("Other"), regardless of causality, is located in the "Reported Adverse Events" section.
Time Frame: 7 days post-vaccination
Population: Solicited Safety Set included all participants who received IP and contributed any solicited AR data.
Measure: Count of Participants; unit: Participants
Groups:
- Part A.1: mRNA-1273.211 50 μg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (COVE), received a single IM booster dose of 50 μg of mRNA-1273.211 on Day 1 of Part A.1.
Arm/Group | Part A.1: mRNA-1273.211 50 μg | Part A.1: mRNA-1273.211 100 μg | Part A.2: mRNA-1273.214 50 μg | Part B: mRNA-1273 100 μg | Part C: mRNA-1273.617.2 50 μg | Part C: mRNA-1273.617.2 100 μg | Part D: mRNA-1273.213 50 μg | Part D: mRNA-1273.213 100 μg | Part E: mRNA-1273.213 100 μg | Part F (Cohort 1): mRNA-1273.529 50 μg | Part F (Cohort 2): mRNA-1273 50 μg | Part F (Cohort 2): mRNA-1273.529 50 μg | Part G: mRNA-1273.214 50 μg | Part H: mRNA-1273.222 50 μg | Part J: mRNA-1273.231 50 μg | Part J: mRNA-1273.815 50 μg
Number analyzed (Participants) | 298 | 591 | 128 | 303 | 577 | 583 | 327 | 583 | 42 | 133 | 350 | 372 | 437 | 507 | 50 | 50
Participants
  Any | 270 | 554 | 113 | 290 | 532 | 548 | 307 | 550 | 41 | 113 | 300 | 323 | 380 | 443 | 44 | 38
  Grade 1 | 140 | 215 | 70 | 95 | 260 | 193 | 134 | 213 | 11 | 59 | 184 | 203 | 220 | 219 | 28 | 23
  Grade 2 | 98 | 250 | 27 | 144 | 201 | 248 | 127 | 227 | 25 | 43 | 88 | 93 | 125 | 165 | 10 | 14
  Grade 3 | 32 | 88 | 16 | 51 | 71 | 107 | 46 | 110 | 5 | 11 | 28 | 27 | 35 | 59 | 6 | 1
  Grade 4 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

2. Primary Outcome: Number of Participants With Unsolicited AEs
Description: An AE was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug related. Any abnormal laboratory test result (hematology, clinical chemistry, or prothrombin time [PT]/partial thromboplastin time [PTT]) or other safety assessment (for example, electrocardiogram, radiological scan, vital sign measurement), including one that worsened from baseline and was considered clinically significant in the medical and scientific judgment of the Investigator was recorded as an AE. Number of participants with unsolicited AEs (SAEs and non-serious AEs) up to 28 days post-vaccination are reported in this outcome measure.
Time Frame: Up to 28 days post-vaccination
Population: Safety Set included all participants who received IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A.1: mRNA-1273.211 50 μg | Part A.1: mRNA-1273.211 100 μg | Part A.2: mRNA-1273.214 50 μg | Part B: mRNA-1273 100 μg | Part C: mRNA-1273.617.2 50 μg | Part C: mRNA-1273.617.2 100 μg | Part D: mRNA-1273.213 50 μg | Part D: mRNA-1273.213 100 μg | Part E: mRNA-1273.213 100 μg | Part F (Cohort 1): mRNA-1273.529 50 μg | Part F (Cohort 2): mRNA-1273 50 μg | Part F (Cohort 2): mRNA-1273.529 50 μg | Part G: mRNA-1273.214 50 μg | Part H: mRNA-1273.222 50 μg | Part J: mRNA-1273.231 50 μg | Part J: mRNA-1273.815 50 μg
Number analyzed (Participants) | 300 | 593 | 135 | 305 | 581 | 586 | 327 | 583 | 42 | 133 | 376 | 375 | 437 | 510 | 50 | 50
Participants | 62 | 126 | 24 | 54 | 134 | 126 | 91 | 135 | 5 | 27 | 80 | 82 | 83 | 119 | 9 | 5

3. Primary Outcome: Number of Participants With SAEs, AEs of Special Interest (AESIs), Medically Attended AEs (MAAEs), and AEs Leading to Study or Treatment Discontinuation
Description: An SAE was defined as any AE that resulted in death, was life-threatening, required inpatient hospitalization or prolongation of existing hospitalization, resulted in disability/permanent damage, was a congenital anomaly/birth defect, or was an important medical event. AESIs included thrombocytopenia, new onset of or worsening of the protocol specified neurologic diseases, anaphylaxis, and myocarditis/pericarditis. An MAAE is an AE that lead to an unscheduled visit to a healthcare practitioner. This included visits to a study site for unscheduled assessments (for example, abnormal laboratory follow-up, and/or coronavirus disease 2019 [COVID-19] and visits to healthcare practitioners external to the study site (for example, urgent care, primary care physician). Number of participants with SAEs, AESIs, MAAEs, and AEs leading to discontinuation up to the end of study (EOS) are reported in this outcome measure.
Time Frame: Day 1 to EOS (Day 366 for Parts A.1, B, C, D, E, and F; and Day 181 for Parts A.2, H, and J)
Population: Safety Set included all participants who received IP.
Measure: Count of Participants; unit: Participants
Arm/Group | Part A.1: mRNA-1273.211 50 μg | Part A.1: mRNA-1273.211 100 μg | Part A.2: mRNA-1273.214 50 μg | Part B: mRNA-1273 100 μg | Part C: mRNA-1273.617.2 50 μg | Part C: mRNA-1273.617.2 100 μg | Part D: mRNA-1273.213 50 μg | Part D: mRNA-1273.213 100 μg | Part E: mRNA-1273.213 100 μg | Part F (Cohort 1): mRNA-1273.529 50 μg | Part F (Cohort 2): mRNA-1273 50 μg | Part F (Cohort 2): mRNA-1273.529 50 μg | Part G: mRNA-1273.214 50 μg | Part H: mRNA-1273.222 50 μg | Part J: mRNA-1273.231 50 μg | Part J: mRNA-1273.815 50 μg
Number analyzed (Participants) | 300 | 593 | 135 | 305 | 581 | 586 | 327 | 583 | 42 | 133 | 376 | 375 | 437 | 510 | 50 | 50
Participants
  SAEs | 6 | 26 | 3 | 15 | 27 | 12 | 8 | 18 | 0 | 2 | 20 | 16 | 23 | 12 | 3 | 2
  AESIs | 3 | 16 | 1 | 14 | 24 | 28 | 6 | 25 | 2 | 2 | 10 | 14 | 19 | 9 | 1 | 2
  MAAEs | 201 | 388 | 58 | 183 | 380 | 417 | 242 | 401 | 34 | 78 | 279 | 271 | 292 | 253 | 27 | 24
  AEs Leading to Discontinuation | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

4. Primary Outcome: Geometric Mean Titer (GMT) of Serum Pseudovirus Neutralizing Antibody (nAb) ID50 Titers Against Omicron BA.1 Variant and Ancestral SARS-CoV-2 at Day 29 - mRNA-1273.214 (50 μg) (Part A.2) Compared to mRNA-1273.211 (50 μg) (Part A.1)
Description: GMT of serum pseudovirus nAb ID50 titers against Omicron BA.1 Variant (B.1.1.529) and ancestral severe acute respiratory syndrome coronavirus (SARS-CoV-2) (D614G) at Day 29 is reported. mRNA-1273.214 (50 μg) as a second booster dose (Part A.2) was compared to mRNA-1273.211 (50 μg) as the first booster dose (Part A.1). Antibody values reported as below the lower limit of quantification (LLOQ) were replaced by 0.5 * LLOQ. Values greater than the upper limit of quantification (ULOQ) were replaced by the ULOQ if actual values were not available. LLOQ was 19.85 arbitrary units (AU)/milliliter (mL) and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Day 29
Population: PPIS-Neg included all participants who received study injection; had pre-booster and Day 29 nAb data; had no major protocol deviations that impacted key or critical data; had no previous human immunodeficiency virus (HIV) infection; and who had no serologic or virologic evidence of SARS-CoV-2 infection at baseline. Overall number of participants analyzed = participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A.2: mRNA-1273.214 50 μg | Part A.1: mRNA-1273.211 50 μg
Number analyzed (Participants) | 76 | 76
titer
  Omicron BA.1 Variant (B.1.1.529) nAb | 4713.5 [3513.5 to 6323.4] | 1897.1 [1433.8 to 2510.1]
  SARS-CoV-2 (D614G) nAb | 5642.3 [4531.1 to 7025.9] | 2861.4 [2396.0 to 3417.1]
Statistical Analysis 1: Comparison: Part A.2: mRNA-1273.214 50 μg vs Part A.1: mRNA-1273.211 50 μg; Test type: Other; Geometric Mean Ratio (GMR) = 2.5, 95% CI 2-sided [2.0 to 3.0] — Omicron BA.1 Variant (B.1.1.529) nAB: Part A.2 versus Part A.1
Statistical Analysis 2: Comparison: Part A.2: mRNA-1273.214 50 μg vs Part A.1: mRNA-1273.211 50 μg; Test type: Other; GMR = 2.0, 95% CI 2-sided [1.7 to 2.3] — SARS-CoV-2 (D614G) nAb: Part A.2 versus Part A.1

5. Primary Outcome: GMT of Serum Pseudovirus nAb ID50 Titers Against Omicron BA.1 Variant and Ancestral SARS-CoV-2 at Day 181 - mRNA-1273.214 (50 μg) (Part A.2) Compared to mRNA-1273.211 (50 μg) (Part A.1)
Description: GMT of serum pseudovirus nAb ID50 titers against Omicron BA.1 Variant (B.1.1.529) and ancestral SARS-CoV-2 (D614G) at Day 181 is reported. mRNA-1273.214 (50 μg) as a second booster dose (Part A.2) was compared to mRNA-1273.211 (50 μg) as the first booster dose (Part A.1). Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available. LLOQ was 19.85 AU/mL and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Day 181
Population: PPIS-Neg included all participants who received study injection; had pre-booster and Day 29 nAb data; had no major protocol deviations that impacted key or critical data; had no previous HIV infection; and who had no serologic or virologic evidence of SARS-CoV-2 infection at baseline. 'Overall number of participants analyzed' = participants evaluable for this outcome measure.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part A.2: mRNA-1273.214 50 μg | Part A.1: mRNA-1273.211 50 μg
Number analyzed (Participants) | 70 | 74
titer
  Omicron BA.1 Variant (B.1.1.529) nAb | 2304.6 [1584.4 to 3352.0] | 379.3 [281.0 to 512.1]
  SARS-CoV-2 (D614G) nAb | 2945.2 [2259.1 to 3839.7] | 1121.4 [927.4 to 1356.1]
Statistical Analysis 1: Comparison: Part A.2: mRNA-1273.214 50 μg vs Part A.1: mRNA-1273.211 50 μg; Test type: Other; Geometric Mean Ratio (GMR) = 6.3, 95% CI 2-sided [4.5 to 8.9] — Omicron BA.1 Variant (B.1.1.529) nAb: Part A.2 versus Part A.1
Statistical Analysis 2: Comparison: Part A.2: mRNA-1273.214 50 μg vs Part A.1: mRNA-1273.211 50 μg; Test type: Other; GMR = 2.8, 95% CI 2-sided [2.1 to 3.6] — SARS-CoV-2 (D614G) nAb: Part A.2 versus Part A.1

6. Primary Outcome: Seroresponse Rate (SRR) (Based on Pre-vaccination Baseline) For Serum Pseudovirus nAb ID50 Titers Against Omicron BA.1 Variant and Ancestral SARS-CoV-2 at Day 29 - mRNA-1273.214 (50 μg) (Part A.2) Compared to mRNA-1273.211 (50 μg) (Part A.1)
Description: Percentage of participants with seroresponse (based on the pre-vaccination baseline) for pseudovirus nAb ID50 against Omicron BA.1 Variant (B.1.1.529) and ancestral SARS-CoV-2 (D614G) at Day 29 are reported. mRNA-1273.214 (50 μg) as a second booster dose (Part A.2) was compared to mRNA-1273.211 (50 μg) as the first booster dose (Part A.1). Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer. LLOQ was 19.85 AU/mL and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A.2: mRNA-1273.214 50 μg | Part A.1: mRNA-1273.211 50 μg
Number analyzed (Participants) | 76 | 76
percentage of participants
  Omicron BA.1 Variant (B.1.1.529) nAb | 100 [95.3 to 100.0] | 98.7 [92.9 to 100.0]
  SARS-CoV-2 (D614G) nAb | 100 [95.3 to 100.0] | 100 [95.3 to 100.0]
Statistical Analysis 1: Comparison: Part A.2: mRNA-1273.214 50 μg vs Part A.1: mRNA-1273.211 50 μg; Test type: Other; Percentage Difference = 1.3, 95% CI 2-sided [-3.1 to 5.6] — Omicron BA.1 Variant (B.1.1.529) nAb: Part A.2 versus Part A.1
Statistical Analysis 2: Comparison: Part A.2: mRNA-1273.214 50 μg vs Part A.1: mRNA-1273.211 50 μg; Test type: Other; Percentage Difference = 0 — SARS-CoV-2 (D614G) nAb: Part A.2 versus Part A.1

7. Primary Outcome: SRR (Based on Pre-booster Baseline) For Serum Pseudovirus nAb ID50 Titers Against Omicron BA.1 Variant and Ancestral SARS-CoV-2 at Day 29 - mRNA-1273.214 (50 μg) (Part A.2) Compared to mRNA-1273.211 (50 μg) (Part A.1)
Description: Percentage of participants with seroresponse (based on the pre-booster baseline) for pseudovirus nAb ID50 against Omicron BA.1 Variant (B.1.1.529) and ancestral SARS-CoV-2 (D614G) at Day 29 are reported. mRNA-1273.214 (50 μg) as a second booster dose (Part A.2) was compared to mRNA-1273.211 (50 μg) as the first booster dose (Part A.1). Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer. LLOQ was 19.85 AU/mL and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Day 29
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A.2: mRNA-1273.214 50 μg | Part A.1: mRNA-1273.211 50 μg
Number analyzed (Participants) | 76 | 76
percentage of participants
  Omicron BA.1 Variant (B.1.1.529) nAb | 97.4 [90.8 to 99.7] | 98.7 [92.9 to 100.0]
  SARS-CoV-2 (D614G) nAb | 93.4 [85.3 to 97.8] | 96.1 [88.9 to 99.2]
Statistical Analysis 1: Comparison: Part A.2: mRNA-1273.214 50 μg vs Part A.1: mRNA-1273.211 50 μg; Test type: Other; Percentage Difference = -1.3, 95% CI 2-sided [-6.9 to 4.3] — Omicron variant (B.1.1.529) nAb: Part A.2 versus Part A.1
Statistical Analysis 2: Comparison: Part A.2: mRNA-1273.214 50 μg vs Part A.1: mRNA-1273.211 50 μg; Test type: Other; Percentage Difference = -2.6, 95% CI 2-sided [-9.6 to 4.5] — SARS-CoV-2 (D614G) nAb: Part A.2 versus Part A.1

8. Primary Outcome: SRR (Based on Pre-vaccination Baseline) For Serum Pseudovirus nAb ID50 Titers Against Omicron BA.1 Variant and Ancestral SARS-CoV-2 at Day 181 - mRNA-1273.214 (50 μg) (Part A.2) Compared to mRNA-1273.211 (50 μg) (Part A.1)
Description: Percentage of participants with seroresponse (based on the pre-vaccination baseline) for pseudovirus nAb ID50 against Omicron BA.1 Variant (B.1.1.529) and ancestral SARS-CoV-2 (D614G) at Day 181 are reported. mRNA-1273.214 (50 μg) as a second booster dose (Part A.2) was compared to mRNA-1273.211 (50 μg) as the first booster dose (Part A.1). Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer. LLOQ was 19.85 AU/mL and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Day 181
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A.2: mRNA-1273.214 50 μg | Part A.1: mRNA-1273.211 50 μg
Number analyzed (Participants) | 70 | 74
percentage of participants
  Omicron BA.1 Variant (B.1.1.529) nAb | 100 [94.9 to 100.0] | 86.5 [76.5 to 93.3]
  SARS-CoV-2 (D614G) nAb | 100 [94.9 to 100.0] | 100 [95.1 to 100.0]
Statistical Analysis 1: Comparison: Part A.2: mRNA-1273.214 50 μg vs Part A.1: mRNA-1273.211 50 μg; Test type: Other; Percentage Difference = 12.9, 95% CI 2-sided [4.1 to 21.6] — Omicron BA.1 variant (B.1.1.529) nAb: Part A.2 versus Part A.1
Statistical Analysis 2: Comparison: Part A.2: mRNA-1273.214 50 μg vs Part A.1: mRNA-1273.211 50 μg; Test type: Other; Percentage Difference = 0 — SARS-CoV-2 (D614G) nAb: Part A.2 versus Part A.1

9. Primary Outcome: SRR (Based on Pre-booster Baseline) For Serum Pseudovirus nAb ID50 Titers Against Omicron BA.1 Variant and Ancestral SARS-CoV-2 at Day 181 - mRNA-1273.214 (50 μg) (Part A.2) Compared to mRNA-1273.211 (50 μg) (Part A.1)
Description: Percentage of participants with seroresponse (based on the pre-booster baseline) for pseudovirus nAb ID50 against Omicron BA.1 Variant (B.1.1.529) and ancestral SARS-CoV-2 (D614G) at Day 181 are reported. mRNA-1273.214 (50 μg) as a second booster dose (Part A.2) was compared to mRNA-1273.211 (50 μg) as the first booster dose (Part A.1). Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer. LLOQ was 19.85 AU/mL and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Day 181
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part A.2: mRNA-1273.214 50 μg | Part A.1: mRNA-1273.211 50 μg
Number analyzed (Participants) | 70 | 74
percentage of participants
  Omicron BA.1 Variant (B.1.1.529) nAb | 81.4 [70.3 to 89.7] | 78.4 [67.3 to 87.1]
  SARS-CoV-2 (D614G) nAb | 71.4 [59.4 to 81.6] | 79.7 [68.8 to 88.2]
Statistical Analysis 1: Comparison: Part A.2: mRNA-1273.214 50 μg vs Part A.1: mRNA-1273.211 50 μg; Test type: Other; Percentage Difference = 2.9, 95% CI 2-sided [-11.4 to 17.1] — Omicron BA.1 variant (B.1.1.529) nAb: Part A.2 versus Part A.1
Statistical Analysis 2: Comparison: Part A.2: mRNA-1273.214 50 μg vs Part A.1: mRNA-1273.211 50 μg; Test type: Other; Percentage Difference = -7.1, 95% CI 2-sided [-21.6 to 7.3] — SARS-CoV-2 (D614G) nAb: Part A.2 versus Part A.1

10. Primary Outcome: GMT of Serum Pseudovirus nAb ID50 Titers Against Omicron BA.1 Variant (B.1.1.529) at Day 29 - Part F (Cohort 2): mRNA-1273.529 and mRNA-1273
Description: GMT of serum pseudovirus nAb ID50 titers against Omicron BA.1 Variant (B.1.1.529) at Day 29 is reported. Part F (Cohort 2) mRNA-1273.529 50 μg was compared to Part F (Cohort 2) mRNA-1273 50 μg. Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available. LLOQ was 19.85 AU/mL and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529.
Time Frame: Day 29
Population: PPIS-Neg included all participants who received study injection; had pre-booster and Day 29 nAb data; had no major protocol deviations that impacted key or critical data; had no previous HIV infection; and who had no serologic or virologic evidence of SARS-CoV-2 infection at baseline.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part F (Cohort 2): mRNA-1273.529 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 273 | 258
titer | 2739.5 [2320.2 to 3234.6] | 1462.1 [1260.1 to 1696.4]
Statistical Analysis 1: Comparison: Part F (Cohort 2): mRNA-1273.529 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; GMR = 1.777, 95% CI 2-sided [1.523 to 2.073] — Omicron BA.1 Variant (B.1.1.529) nAb - Part F (Cohort 2): mRNA-1273.529 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg

11. Primary Outcome: SRR (Based on Pre-vaccination Baseline) for Serum Pseudovirus nAb ID50 Titers Against Omicron BA.1 Variant (B.1.1.529) at Day 29 - Part F (Cohort 2): mRNA-1273.529 and mRNA-1273
Description: Percentage of participants with seroresponse (based on the pre-vaccination baseline) for pseudovirus nAb ID50 against Omicron BA.1 Variant (B.1.1.529) at Day 29 are reported. Part F (Cohort 2) mRNA-1273.529 50 μg was compared to Part F (Cohort 2) mRNA-1273 50 μg. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 19.85 AU/mL and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529.
Time Frame: Day 29
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part F (Cohort 2): mRNA-1273.529 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 273 | 258
percentage of participants | 99.6 [98.0 to 100.0] | 99.2 [97.2 to 99.9]
Statistical Analysis 1: Comparison: Part F (Cohort 2): mRNA-1273.529 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; Percentage Difference = 0.6, 95% CI 2-sided [-1.7 to 3.0] — Omicron BA.1 Variant (B.1.1.529) nAb - Part F (Cohort 2): mRNA-1273.529 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg

12. Primary Outcome: SRR (Based on Pre-booster Baseline) for Serum Pseudovirus nAb ID50 Titers Against Omicron BA.1 Variant (B.1.1.529) at Day 29 - Part F (Cohort 2): mRNA-1273.529 and mRNA-1273
Description: Percentage of participants with seroresponse (based on the pre-booster baseline) for pseudovirus nAb ID50 against Omicron BA.1 Variant (B.1.1.529) at Day 29 are reported. Part F (Cohort 2) mRNA-1273.529 50 μg was compared to Part F (Cohort 2) mRNA-1273 50 μg. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 19.85 AU/mL and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529.
Time Frame: Day 29
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part F (Cohort 2): mRNA-1273.529 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 273 | 258
percentage of participants | 71.4 [65.7 to 76.7] | 53.5 [47.2 to 59.7]
Statistical Analysis 1: Comparison: Part F (Cohort 2): mRNA-1273.529 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; Percentage Difference = 17.9, 95% CI 2-sided [9.8 to 26.0] — Omicron BA.1 Variant (B.1.1.529) nAb - Part F (Cohort 2): mRNA-1273.529 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg

13. Primary Outcome: GMT of Serum Pseudovirus nAb ID50 Titers Against Omicron BA.1 Variant (B.1.1.529) and Ancestral SARS-CoV-2 (D614G) at Day 29 - mRNA-1273.214 (Part G) Compared to mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273)
Description: GMT of serum pseudovirus nAb ID50 titers against Omicron BA.1 Variant (B.1.1.529) and ancestral SARS-CoV-2 (D614G) at Day 29 is reported. mRNA-1273.214 (Part G) was compared the mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273). Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available. LLOQ was 19.85 AU/mL and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Day 29
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part G: mRNA-1273.214 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 334 | 258
titer
  Omicron BA.1 Variant (B.1.1.529) nAb | 2370.5 [2068.8 to 2716.1] | 1462.1 [1260.1 to 1696.4]
  SARS-CoV-2 (D614G) nAb | 5971.6 [5316.7 to 6707.2] | 5621.4 [5029.2 to 6283.4]
Statistical Analysis 1: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; GMR = 1.744, 97.5% CI 2-sided [1.492 to 2.040] — Omicron BA.1 Variant (B.1.1.529) nAb: Part G: mRNA-1273.214 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg
Statistical Analysis 2: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; GMR = 1.211, 97.5% CI 2-sided [1.074 to 1.366] — SARS-CoV-2 (D614G) nAb: Part G: mRNA-1273.214 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg

14. Primary Outcome: GMT of Serum Pseudovirus nAb ID50 Titers Against Omicron BA.1 Variant (B.1.1.529) and Ancestral SARS-CoV-2 (D614G) at Day 91 - mRNA-1273.214 (Part G) Compared to mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273)
Description: GMT of serum pseudovirus nAb ID50 titers against Omicron BA.1 Variant (B.1.1.529) and ancestral SARS-CoV-2 (D614G) at Day 91 is reported. mRNA-1273.214 (Part G) was compared the mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273). Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available. LLOQ was 19.85 AU/mL and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Day 91
Population: as for outcome 5
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part G: mRNA-1273.214 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 329 | 243
titer
  Omicron BA.1 Variant (B.1.1.529) nAb | 967.3 [835.0 to 1120.6] | 624.2 [533.1 to 730.9]
  SARS-CoV-2 (D614G) nAb | 3431.5 [3066.7 to 3839.8] | 3447.1 [3054.7 to 3889.9]
Statistical Analysis 1: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; GMR = 1.676, 97.5% CI 2-sided [1.396 to 2.013] — Omicron BA.1 Variant (B.1.1.529) nAb: Part G: mRNA-1273.214 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg
Statistical Analysis 2: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; GMR = 1.105, 97.5% CI 2-sided [0.970 to 1.260] — SARS-CoV-2 (D614G) nAb: Part G: mRNA-1273.214 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg

15. Primary Outcome: SRR (Based on the Pre-vaccination Baseline) for Serum Pseudovirus nAb ID50 Titers Against Omicron BA.1 Variant (B.1.1.529) at Day 29 - mRNA-1273.214 (Part G) Compared to mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273)
Description: Percentage of participants with seroresponse (based on the pre-vaccination baseline) for pseudovirus nAb ID50 against Omicron BA.1 Variant (B.1.1.529) at Day 29 are reported. mRNA-1273.214 (Part G) was compared the mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273). Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer. LLOQ was 19.85 AU/mL and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529.
Time Frame: Day 29
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part G: mRNA-1273.214 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 334 | 258
percentage of participants | 100 [98.9 to 100.0] | 99.2 [97.2 to 99.9]
Statistical Analysis 1: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; Percentage Difference = 1.5, 97.5% CI 2-sided [-1.1 to 4.1] — Omicron BA.1 Variant (B.1.1.529) nAb: Part G: mRNA-1273.214 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg

16. Primary Outcome: SRR (Based on the Pre-booster Baseline) for Serum Pseudovirus nAb ID50 Titers Against Omicron BA.1 Variant (B.1.1.529) at Day 29 - mRNA-1273.214 (Part G) Compared to mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273)
Description: Percentage of participants with seroresponse (based on the pre-booster baseline) for pseudovirus nAb ID50 against Omicron BA.1 Variant (B.1.1.529) at Day 29 are reported. mRNA-1273.214 (Part G) was compared the mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273). Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 19.85 AU/mL and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529.
Time Frame: Day 29
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part G: mRNA-1273.214 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 334 | 258
percentage of participants | 75.1 [70.2 to 79.7] | 53.5 [47.2 to 59.7]
Statistical Analysis 1: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; Percentage Difference = 21.5, 97.5% CI 2-sided [12.8 to 30.2] — Omicron BA.1 Variant (B.1.1.529) nAb: Part G: mRNA-1273.214 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg

17. Primary Outcome: SRR (Based on the Pre-vaccination Baseline) for Serum Pseudovirus nAb ID50 Titers Against Omicron BA.1 Variant (B.1.1.529) at Day 91 - mRNA-1273.214 (Part G) Compared to mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273)
Description: Percentage of participants with seroresponse (based on the pre-vaccination baseline) for pseudovirus nAb ID50 against Omicron BA.1 Variant (B.1.1.529) at Day 91 are reported. mRNA-1273.214 (Part G) was compared the mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273). Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 19.85 AU/mL and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529.
Time Frame: Day 91
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part G: mRNA-1273.214 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 329 | 243
percentage of participants | 98.2 [96.1 to 99.3] | 96.3 [93.0 to 98.3]
Statistical Analysis 1: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; Percentage Difference = 1.8, 97.5% CI 2-sided [-1.9 to 5.6] — Omicron BA.1 Variant (B.1.1.529) nAb: Part G: mRNA-1273.214 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg

18. Primary Outcome: SRR (Based on the Pre-booster Baseline) for Serum Pseudovirus nAb ID50 Titers Against Omicron BA.1 Variant (B.1.1.529) at Day 91 - mRNA-1273.214 (Part G) Compared to mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273)
Description: Percentage of participants with seroresponse (based on the pre-booster baseline) for pseudovirus nAb ID50 against Omicron BA.1 Variant (B.1.1.529) at Day 91 are reported. mRNA-1273.214 (Part G) was compared the mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273). Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 19.85 AU/mL and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529.
Time Frame: Day 91
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part G: mRNA-1273.214 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 329 | 243
percentage of participants | 38.6 [33.3 to 44.1] | 17.7 [13.1 to 23.1]
Statistical Analysis 1: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; Percentage Difference = 20.6, 97.5% CI 2-sided [12.4 to 28.7] — Omicron BA.1 Variant (B.1.1.529) nAb: Part G: mRNA-1273.214 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg

19. Primary Outcome: GMT of Serum Pseudovirus nAb ID50 Titers Against Omicron BA.4/BA.5 Variant and Ancestral SARS-CoV-2 (D614G) at Day 29 - mRNA-1273.222 (Part H) Compared to mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273)
Description: GMT of serum pseudovirus nAb ID50 titers against BA.4/BA.5 and ancestral SARS-CoV-2 (D614G) at Day 29 is reported. mRNA-1273.222 (Part H) was compared to mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273). Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available. LLOQ was 36.7 AU/mL and ULOQ was 13705 AU/mL for ID50 titer against BA.4/BA.5. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Day 29
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part H: mRNA-1273.222 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 209 | 258
titer
  Omicron Variant (BA.4/BA.5) | 2322.6 [1919.9 to 2809.7] | 483.0 [423.1 to 551.3]
  SARS-CoV-2 (D614G) nAb | 7328.4 [6390.6 to 8403.8] | 5621.4 [5029.2 to 6283.4]
Statistical Analysis 1: Comparison: Part H: mRNA-1273.222 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; GMR = 6.412, 95% CI 2-sided [5.369 to 7.658] — Omicron Variant (BA.4/BA.5) nAb: Part H mRNA-1273.222 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg
Statistical Analysis 2: Comparison: Part H: mRNA-1273.222 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; GMR = 1.967, 95% CI 2-sided [1.708 to 2.265] — SARS-CoV-2 (D614G) nAb: Part H mRNA-1273.222 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg

20. Primary Outcome: SRR (Based on Pre-vaccination Baseline) for Serum Pseudovirus nAb ID50 Titers Against Omicron BA.4/BA.5 Variant and Ancestral SARS-CoV-2 (D614G) at Day 29 - mRNA-1273.222 (Part H) Compared to mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273)
Description: Percentage of participants with seroresponse (based on the pre-vaccination baseline) for pseudovirus nAb ID50 against BA.4/BA.5 and ancestral SARS-CoV-2 (D614G) at Day 29 are reported. mRNA-1273.222 (Part H) was compared to mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273). Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 36.7 AU/mL and ULOQ was 13705 AU/mL for ID50 titer against BA.4/BA.5. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Day 29
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part H: mRNA-1273.222 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 209 | 258
percentage of participants
  Omicron Variant (BA.4/BA.5) | 98.1 [95.2 to 99.5] | 86.3 [81.5 to 90.3]
  SARS-CoV-2 (D614G) nAb | 100 [98.3 to 100.0] | 100 [98.6 to 100.0]
Statistical Analysis 1: Comparison: Part H: mRNA-1273.222 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; Percentage Difference = 12.2, 95% CI 2-sided [6.9 to 17.4] — Omicron Variant (BA.4/BA.5) nAb: Part H mRNA-1273.222 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg
Statistical Analysis 2: Comparison: Part H: mRNA-1273.222 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; Percentage Difference = 0 — SARS-CoV-2 (D614G) nAb: Part H mRNA-1273.222 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg

21. Primary Outcome: SRR (Based on Pre-booster Baseline) for Serum Pseudovirus nAb ID50 Titers Against Omicron BA.4/BA.5 Variant and Ancestral SARS-CoV-2 (D614G) at Day 29 - mRNA-1273.222 (Part H) Compared to mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273)
Description: Percentage of participants with seroresponse (based on the pre-booster baseline) for pseudovirus nAb ID50 against BA.4/BA.5 and ancestral SARS-CoV-2 (D614G) at Day 29 are reported. mRNA-1273.222 (Part H) was compared to mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273). Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 36.7 AU/mL and ULOQ was 13705 AU/mL for ID50 titer against BA.4/BA.5. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Day 29
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part H: mRNA-1273.222 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 209 | 258
percentage of participants
  Omicron Variant (BA.4/BA.5) | 91.4 [86.7 to 94.8] | 37.6 [31.7 to 43.8]
  SARS-CoV-2 (D614G) nAb | 80.9 [74.9 to 86.0] | 43.0 [36.9 to 49.3]
Statistical Analysis 1: Comparison: Part H: mRNA-1273.222 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; Percentage Difference = 54.7, 95% CI 2-sided [47.5 to 61.8] — Omicron Variant (BA.4/BA.5) nAb: Part H mRNA-1273.222 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg
Statistical Analysis 2: Comparison: Part H: mRNA-1273.222 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; Percentage Difference = 37.6, 95% CI 2-sided [29.3 to 45.9] — SARS-CoV-2 (D614G) nAb: Part H mRNA-1273.222 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg

22. Primary Outcome: GMT of Serum Pseudovirus nAb ID50 Titers Against SARS-CoV-2 XBB.1.5, BA.4/BA.5, and SARS-CoV-2 BQ.1.1 at Day 15 - Part J: mRNA-1273.231 and mRNA-1273.815
Description: GMT of serum pseudovirus nAb ID50 titers against SARS-CoV-2 XBB.1.5, BA.4/BA.5, and SARS-CoV-2 BQ.1.1 at Day 15 is reported. Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available. Antibody values reported as below the lower limit of detection (LOD) are replaced by 0.5 * LOD. LOD was 10 AU/mL for ID50 titer against XBB.1.5 and BQ.1.1. LLOQ was 36.7 AU/mL and ULOQ was 13705 AU/mL for ID50 titer against BA.4/BA.5.
Time Frame: Day 15
Population: PPIS included all participants who received study injection; had pre-booster and Day 15 nAb data; and who had no major protocol deviations that impacted key or critical data.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Groups:
- Part J: mRNA-1273.231 50 μg: Participants who previously received a primary series of mRNA vaccine, a first booster dose of a monovalent mRNA vaccine, and a second booster dose of a bivalent mRNA vaccine against SARS-CoV-2, received a third IM booster dose of 50 ug of mRNA-1273.231 on Day 1 of Part J.
Arm/Group | Part J: mRNA-1273.231 50 μg | Part J: mRNA-1273.815 50 μg
Number analyzed (Participants) | 49 | 49
titer
  SARS-CoV-2 (XBB.1.5) nAb | 1751.2 [1212.5 to 2529.4] | 2579.0 [1809.1 to 3676.7]
  SARS-CoV-2 (BA.4/BA.5) nAb | 9600.1 [7392.8 to 12466.4] | 9673.4 [6965.6 to 13433.8]
  SARS-CoV-2 (BQ.1.1) nAb | 1806.7 [1294.1 to 2522.2] | 1894.1 [1383.2 to 2593.6]

23. Primary Outcome: GMT of Serum Pseudovirus nAb ID50 Titers Against SARS-CoV-2 XBB.1.5, BA.4/BA.5, and SARS-CoV-2 BQ.1.1 at Day 29 - Part J: mRNA-1273.231 and mRNA-1273.815
Description: GMT of serum pseudovirus nAb ID50 titers against SARS-CoV-2 XBB.1.5, BA.4/BA.5, and SARS-CoV-2 BQ.1.1 at Day 29 is reported. Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available. Antibody values reported as below the LOD are replaced by 0.5 * LOD. LOD was 10 AU/mL for ID50 titer against XBB.1.5 and BQ.1.1. LLOQ was 36.7 AU/mL and ULOQ was 13705 AU/mL for ID50 titer against BA.4/BA.5.
Time Frame: Day 29
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part J: mRNA-1273.231 50 μg | Part J: mRNA-1273.815 50 μg
Number analyzed (Participants) | 49 | 49
titer
  SARS-CoV-2 (XBB.1.5) nAb | 1985.5 [1388.7 to 2838.8] | 2710.6 [1778.3 to 4131.8]
  SARS-CoV-2 (BA.4/BA.5) nAb | 10469.7 [7771.5 to 14104.8] | 11231.0 [7883.5 to 15999.9]
  SARS-CoV-2 (BQ.1.1) nAb | 1727.4 [1293.0 to 2307.6] | 1991.1 [1308.6 to 3029.5]

24. Primary Outcome: Geometric Mean Fold Rise (GMFR) of Serum Pseudovirus nAb ID50 Titers Against SARS-CoV-2 XBB.1.5, BA.4/BA.5, and SARS-CoV-2 BQ.1.1 at Day 15 - Part J: mRNA-1273.231 and mRNA-1273.815
Description: GMFR of serum pseudovirus nAb ID50 titers against SARS-CoV-2 XBB.1.5, BA.4/BA.5, and SARS-CoV-2 BQ.1.1 at Day 15 is reported. GMFR measures the changes in immunogenicity titers or levels from Baseline within participants. Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available. Antibody values reported as below the LOD are replaced by 0.5 * LOD. LOD was 10 AU/mL for ID50 titer against XBB.1.5 and BQ.1.1. LLOQ was 36.7 AU/mL and ULOQ was 13705 AU/mL for ID50 titer against BA.4/BA.5.
Time Frame: Day 15
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part J: mRNA-1273.231 50 μg | Part J: mRNA-1273.815 50 μg
Number analyzed (Participants) | 49 | 49
ratio
  SARS-CoV-2 (XBB.1.5) nAb | 11.0 [8.4 to 14.5] | 16.7 [12.8 to 21.7]
  SARS-CoV-2 (BA.4/BA.5) nAb | 5.0 [3.8 to 6.6] | 6.3 [4.8 to 8.2]
  SARS-CoV-2 (BQ.1.1) nAb | 5.7 [4.5 to 7.2] | 5.9 [4.8 to 7.4]

25. Primary Outcome: GMFR of Serum Pseudovirus nAb ID50 Titers Against SARS-CoV-2 XBB.1.5, BA.4/BA.5, and SARS-CoV-2 BQ.1.1 at Day 29 - Part J: mRNA-1273.231 and mRNA-1273.815
Description: GMFR of serum pseudovirus nAb ID50 titers against SARS-CoV-2 XBB.1.5, BA.4/BA.5, and SARS-CoV-2 BQ.1.1 at Day 29 is reported. GMFR measures the changes in immunogenicity titers or levels from Baseline within participants. Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available. Antibody values reported as below the LOD are replaced by 0.5 * LOD. LOD was 10 AU/mL for ID50 titer against XBB.1.5 and BQ.1.1. LLOQ was 36.7 AU/mL and ULOQ was 13705 AU/mL for ID50 titer against BA.4/BA.5
Time Frame: Day 29
Population: as for outcome 22
Measure: Geometric Mean (95% Confidence Interval); unit: ratio
Arm/Group | Part J: mRNA-1273.231 50 μg | Part J: mRNA-1273.815 50 μg
Number analyzed (Participants) | 49 | 49
ratio
  SARS-CoV-2 (XBB.1.5) nAb | 12.5 [9.6 to 16.3] | 17.5 [13.0 to 23.6]
  SARS-CoV-2 (BA.4/BA.5) nAb | 5.5 [4.2 to 7.1] | 7.3 [5.4 to 9.9]
  SARS-CoV-2 (BQ.1.1) nAb | 5.4 [4.3 to 7.0] | 6.2 [4.6 to 8.4]

26. Primary Outcome: SRR (Based on the Pre-vaccination Baseline) for Serum Pseudovirus nAb ID50 Titers Against BA.4/BA.5 at Day 15 - Part J: mRNA-1273.231 and mRNA-1273.815
Description: Percentage of participants with seroresponse (based on the pre-vaccination baseline) for pseudovirus nAb ID50 against BA.4/BA.5 at Day 15 are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 36.7 AU/mL and ULOQ was 13705 AU/mL for ID50 titer against BA.4/BA.5.
Time Frame: Day 15
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part J: mRNA-1273.231 50 μg | Part J: mRNA-1273.815 50 μg
Number analyzed (Participants) | 49 | 49
percentage of participants | 100 [88.8 to 100.0] | 100 [90.5 to 100.0]

27. Primary Outcome: SRR (Based on the Pre-booster Baseline) for Serum Pseudovirus nAb ID50 Titers Against BA.4/BA.5 at Day 15 - Part J: mRNA-1273.231 and mRNA-1273.815
Description: Percentage of participants with seroresponse (based on the pre-booster baseline) for pseudovirus nAb ID50 against BA.4/BA.5 at Day 15 are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 36.7 AU/mL and ULOQ was 13705 AU/mL for ID50 titer against BA.4/BA.5.
Time Frame: Day 15
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part J: mRNA-1273.231 50 μg | Part J: mRNA-1273.815 50 μg
Number analyzed (Participants) | 49 | 49
percentage of participants | 61.2 [46.2 to 74.8] | 69.4 [54.6 to 81.7]

28. Primary Outcome: SRR (Based on the Pre-vaccination Baseline) for Serum Pseudovirus nAb ID50 Titers Against BA.4/BA.5 at Day 29 - Part J: mRNA-1273.231 and mRNA-1273.815
Description: Percentage of participants with seroresponse (based on the pre-vaccination baseline) for pseudovirus nAb ID50 against BA.4/BA.5 at Day 29 are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 36.7 AU/mL and ULOQ was 13705 AU/mL for ID50 titer against BA.4/BA.5.
Time Frame: Day 29
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part J: mRNA-1273.231 50 μg | Part J: mRNA-1273.815 50 μg
Number analyzed (Participants) | 49 | 49
percentage of participants | 100 [88.8 to 100.0] | 100 [90.5 to 100.0]

29. Primary Outcome: SRR (Based on the Pre-booster Baseline) for Serum Pseudovirus nAb ID50 Titers Against BA.4/BA.5 at Day 29 - Part J: mRNA-1273.231 and mRNA-1273.815
Description: Percentage of participants with seroresponse (based on the pre-booster baseline) for pseudovirus nAb ID50 against BA.4/BA.5 at Day 29 are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 36.7 AU/mL and ULOQ was 13705 AU/mL for ID50 titer against BA.4/BA.5.
Time Frame: Day 29
Population: as for outcome 22
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part J: mRNA-1273.231 50 μg | Part J: mRNA-1273.815 50 μg
Number analyzed (Participants) | 49 | 49
percentage of participants | 61.2 [46.2 to 74.8] | 67.3 [52.5 to 80.1]

30. Secondary Outcome: GMT of Serum Pseudovirus nAb ID50 Titers Against Ancestral SARS-CoV-2 (D614G) at Day 29 - Part F (Cohort 2): mRNA-1273.529 and mRNA-1273
Description: GMT of serum pseudovirus nAb ID50 titers against ancestral SARS-CoV-2 (D614G) at Day 29 is reported. Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Day 29
Population: as for outcome 10
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part F (Cohort 2): mRNA-1273.529 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 273 | 258
titer | 4951.8 [4349.0 to 5638.0] | 5621.4 [5029.2 to 6283.4]
Statistical Analysis 1: Comparison: Part F (Cohort 2): mRNA-1273.529 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; GMR = 0.836, 95% CI 2-sided [0.745 to 0.938] — SARS-CoV-2 (D614G) nAb: Part F (Cohort 2): mRNA-1273.529 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg

31. Secondary Outcome: SRR (Based on the Pre-vaccination Baseline) for Serum Pseudovirus nAb ID50 Titers Against Ancestral SARS-CoV-2 (D614G) at Day 29 - Part F (Cohort 2): mRNA-1273.529 and mRNA-1273
Description: Percentage of participants with seroresponse (based on the pre-vaccination baseline) for pseudovirus nAb ID50 against ancestral SARS-CoV-2 (D614G) at Day 29 are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Day 29
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part F (Cohort 2): mRNA-1273.529 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 273 | 258
percentage of participants | 100 [98.7 to 100] | 100 [98.6 to 100]
Statistical Analysis 1: Comparison: Part F (Cohort 2): mRNA-1273.529 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; SRR Difference = 0 — SARS-CoV-2 (D614G) nAb: Part F (Cohort 2): mRNA-1273.529 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg 95% CI could not be calculated due to the SRR difference is 0

32. Secondary Outcome: SRR (Based on the Pre-booster Baseline) for Serum Pseudovirus nAb ID50 Titers Against Ancestral SARS-CoV-2 (D614G) at Day 29 - Part F (Cohort 2): mRNA-1273.529 and mRNA-1273
Description: Percentage of participants with seroresponse (based on the pre-booster baseline) for pseudovirus nAb ID50 against ancestral SARS-CoV-2 (D614G) at Day 29 are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Day 29
Population: as for outcome 10
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part F (Cohort 2): mRNA-1273.529 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 273 | 258
percentage of participants | 29.7 [24.3 to 35.5] | 43.0 [36.9 to 49.3]
Statistical Analysis 1: Comparison: Part F (Cohort 2): mRNA-1273.529 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; SRR Difference = -13.1, 95% CI 2-sided [-21.2 to -5.0] — SARS-CoV-2 (D614G) nAb: Part F (Cohort 2): mRNA-1273.529 50 μg versus Part F (Cohort 2): mRNA-1273 50 μg

33. Secondary Outcome: SRR (Based on the Pre-vaccination Baseline) for Serum Pseudovirus nAb ID50 Titers Against Ancestral SARS-CoV-2 (D614G) on Days 29, 91, 181, and 366 - mRNA-1273.214 (Part G) and mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273)
Description: Percentage of participants with seroresponse (based on the pre-vaccination baseline) for pseudovirus nAb ID50 against ancestral SARS-CoV-2 (D614G) on Days 29, 91, 181, and 366 are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Days 29, 91, 181, and 366
Population: PPIS-Neg included all participants who received study injection; had pre-booster and Day 29 nAb data; had no major protocol deviations that impacted key or critical data; had no previous HIV infection; and who had no serologic or virologic evidence of SARS-CoV-2 infection at baseline. 'Number analyzed' = participants evaluable at specified timepoints.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part G: mRNA-1273.214 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 334 | 258
percentage of participants
  Day 29 | 100 [98.9 to 100.0] | 100 [98.6 to 100.0]
  Day 91: number analyzed (Participants) | 329 | 243
  Day 91 | 100 [98.9 to 100.0] | 99.6 [97.7 to 100.0]
  Day 181: number analyzed (Participants) | 308 | 239
  Day 181 | 99.4 [97.7 to 99.9] | 99.6 [97.7 to 100.0]
  Day 366: number analyzed (Participants) | 193 | 179
  Day 366 | 97.9 [94.8 to 99.4] | 99.4 [96.9 to 100.0]
Statistical Analysis 1: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; SRR Difference = 0 — SARS-CoV-2 (D614G) nAb at Day 29: Part G versus Part F (Cohort 2) mRNA-1273 95% CI could not be calculated due to the SRR difference is 0
Statistical Analysis 2: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; SRR Difference = 0.9, 97.5% CI 2-sided [-1.6 to 3.5] — SARS-CoV-2 (D614G) nAb at Day 91: Part G versus Part F (Cohort 2) mRNA-1273
Statistical Analysis 3: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; SRR Difference = -0.1, 95% CI 2-sided [-2.3 to 2.1] — SARS-CoV-2 (D614G) nAb at Day 181: Part G versus Part F (Cohort 2) mRNA-1273
Statistical Analysis 4: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; SRR Difference = -1.9, 95% CI 2-sided [-5.3 to 1.5] — SARS-CoV-2 (D614G) nAb at Day 366: Part G versus Part F (Cohort 2) mRNA-1273

34. Secondary Outcome: SRR (Based on the Pre-booster Baseline) for Serum Pseudovirus nAb ID50 Titers Against Ancestral SARS-CoV-2 (D614G) on Days 29, 91, 181, and 366 - mRNA-1273.214 (Part G) and mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273)
Description: Percentage of participants with seroresponse (based on the pre-booster baseline) for pseudovirus nAb ID50 against ancestral SARS-CoV-2 (D614G) on Days 29, 91, 181, and 366 are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Days 29, 91, 181, and 366
Population: as for outcome 33
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part G: mRNA-1273.214 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 334 | 258
percentage of participants
  Day 29 | 53.9 [48.4 to 59.3] | 43.0 [36.9 to 49.3]
  Day 91: number analyzed (Participants) | 329 | 243
  Day 91 | 27.4 [22.6 to 32.5] | 18.1 [13.5 to 23.5]
  Day 181: number analyzed (Participants) | 308 | 239
  Day 181 | 29.5 [24.5 to 35.0] | 19.2 [14.4 to 24.8]
  Day 366: number analyzed (Participants) | 193 | 179
  Day 366 | 32.6 [26.1 to 39.7] | 27.9 [21.5 to 35.1]
Statistical Analysis 1: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; SRR Difference = 10.9, 97.5% CI 2-sided [1.7 to 20.1] — SARS-CoV-2 (D614G) nAb at Day 29: Part G versus Part F (Cohort 2) mRNA-1273
Statistical Analysis 2: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; SRR Difference = 9.2, 97.5% CI 2-sided [1.4 to 17.0] — SARS-CoV-2 (D614G) nAb at Day 91: Part G versus Part F (Cohort 2) mRNA-1273
Statistical Analysis 3: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; SRR Difference = 10.1, 95% CI 2-sided [3.0 to 17.2] — SARS-CoV-2 (D614G) nAb at Day 181: Part G versus Part F (Cohort 2) mRNA-1273
Statistical Analysis 4: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; SRR Difference = 4.3, 95% CI 2-sided [-5.0 to 13.6] — SARS-CoV-2 (D614G) nAb at Day 366: Part G versus Part F (Cohort 2) mRNA-1273

35. Secondary Outcome: GMT of Serum Pseudovirus nAb ID50 Titers Against BA.4/BA.5 at Day 181 - mRNA-1273.222 (Part H)
Description: GMT of serum pseudovirus nAb ID50 titers against BA.4/BA.5 at Day 181 is reported. Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available. LLOQ was 36.7 AU/mL and ULOQ was 13705 AU/mL for ID50 titer against BA.4/BA.5.
Time Frame: Day 181
Population: PPIS-Neg included all participants who received study injection; had pre-booster and Day 29 nAb data; had no major protocol deviations that impacted key or critical data; had no previous HIV infection; and who had no serologic or virologic evidence of SARS-CoV-2 infection at baseline. 'Overall number of participants analyzed' = participants evaluable for this endpoint.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part H: mRNA-1273.222 50 μg
Number analyzed (Participants) | 189
titer | 1424.7 [1123.5 to 1806.7]

36. Secondary Outcome: GMT of Serum Pseudovirus nAb ID50 Titers Against Ancestral SARS-CoV-2 (D614G) at Day 181 - mRNA-1273.222 (Part H) and mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273)
Description: GMT of serum pseudovirus nAb ID50 titers against ancestral SARS-CoV-2 (D614G) at Day 181 is reported. Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Day 181
Population: as for outcome 35
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part H: mRNA-1273.222 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 189 | 239
titer | 2906.6 [2465.4 to 3426.9] | 2393.3 [2047.4 to 2797.6]
Statistical Analysis 1: Comparison: Part H: mRNA-1273.222 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; GMR = 1.818, 95% CI 2-sided [1.469 to 2.249] — SARS-CoV-2 (D614G) nAb: Part H versus Part F (Cohort 2) mRNA-1273

37. Secondary Outcome: SRR (Based on Pre-vaccination Baseline) for Serum Pseudovirus nAb ID50 Titers Against BA.4/BA.5 at Day 181 - mRNA-1273.222 (Part H)
Description: Percentage of participants with seroresponse (based on the pre-vaccination baseline) for pseudovirus nAb ID50 against BA.4/BA.5 at Day 181 are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 36.7 AU/mL and ULOQ was 13705 AU/mL for ID50 titer against BA.4/BA.5.
Time Frame: Day 181
Population: as for outcome 35
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part H: mRNA-1273.222 50 μg
Number analyzed (Participants) | 189
percentage of participants | 89.9 [84.7 to 93.8]

38. Secondary Outcome: SRR (Based on Pre-vaccination Baseline) for Serum Pseudovirus nAb ID50 Titers Against Ancestral SARS-CoV-2 (D614G) at Day 181 - mRNA-1273.222 (Part H) and mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273)
Description: Percentage of participants with seroresponse (based on the pre-vaccination baseline) for pseudovirus nAb ID50 against ancestral SARS-CoV-2 (D614G) at Day 181 are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Day 181
Population: as for outcome 35
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part H: mRNA-1273.222 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 189 | 239
percentage of participants | 100 [98.1 to 100.0] | 99.6 [97.7 to 100.0]
Statistical Analysis 1: Comparison: Part H: mRNA-1273.222 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; SRR Difference = 0, 95% CI 2-sided [-2.6 to 2.5] — SARS-CoV-2 (D614G) nAb: Part H versus Part F (Cohort 2) mRNA-1273

39. Secondary Outcome: SRR (Based on Pre-booster Baseline) for Serum Pseudovirus nAb ID50 Titers Against BA.4/BA.5 at Day 181 - mRNA-1273.222 (Part H)
Description: Percentage of participants with seroresponse (based on the pre-booster baseline) for pseudovirus nAb ID50 against BA.4/BA.5 at Day 181 are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 36.7 AU/mL and ULOQ was 13705 AU/mL for ID50 titer against BA.4/BA.5.
Time Frame: Day 181
Population: as for outcome 35
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part H: mRNA-1273.222 50 μg
Number analyzed (Participants) | 189
percentage of participants | 77.2 [70.6 to 83.0]

40. Secondary Outcome: SRR (Based on Pre-booster Baseline) for Serum Pseudovirus nAb ID50 Titers Against Ancestral SARS-CoV-2 (D614G) at Day 181 - mRNA-1273.222 (Part H) and mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273)
Description: Percentage of participants with seroresponse (based on the pre-booster baseline) for pseudovirus nAb ID50 against ancestral SARS-CoV-2 (D614G) at Day 181 are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Day 181
Population: as for outcome 35
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part H: mRNA-1273.222 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 189 | 239
percentage of participants | 45.0 [37.7 to 52.4] | 19.2 [14.4 to 24.8]
Statistical Analysis 1: Comparison: Part H: mRNA-1273.222 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; SRR Difference = 25.5, 95% CI 2-sided [16.9 to 34.1] — SARS-CoV-2 (D614G) nAb: Part H versus Part F (Cohort 2) mRNA-1273

41. Secondary Outcome: SRR (Based on the Pre-vaccination Baseline) for Serum Pseudovirus nAb ID50 Titers Against Omicron BA.1 Variant (B.1.1.529) at Days 181 and 366 - mRNA-1273.214 (Part G) and mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273)
Description: Percentage of participants with seroresponse (based on the pre-vaccination baseline) for pseudovirus nAb ID50 against Omicron BA.1 Variant (B.1.1.529) at Days 181 and 366 are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 19.85 AU/mL and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529.
Time Frame: Days 181 and 366
Population: PPIS-Neg included all participants who received study injection; had pre-booster and Day 29 nAb data; had no major protocol deviations that impacted key or critical data; had no previous HIV infection; and who had no serologic or virologic evidence of SARS-CoV-2 infection at baseline. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable at specified timepoint.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part G: mRNA-1273.214 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 308 | 239
percentage of participants
  Day 181 | 94.5 [91.3 to 96.7] | 90.3 [85.8 to 93.7]
  Day 366: number analyzed (Participants) | 193 | 179
  Day 366 | 94.8 [90.6 to 97.5] | 89.8 [84.4 to 93.9]
Statistical Analysis 1: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; SRR Difference = 5.0, 95% CI 2-sided [0.3 to 9.8] — Omicron BA.1 Variant (B.1.1.529) nAb at Day 181: Part G versus Part F (Cohort 2) mRNA-1273
Statistical Analysis 2: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; SRR Difference = 5.6, 95% CI 2-sided [-0.3 to 11.5] — Omicron BA.1 Variant (B.1.1.529) nAb at Day 366: Part G versus Part F (Cohort 2) mRNA-1273

42. Secondary Outcome: SRR (Based on the Pre-booster Baseline) for Serum Pseudovirus nAb ID50 Titers Against Omicron BA.1 Variant (B.1.1.529) at Days 181 and 366 - mRNA-1273.214 (Part G) and mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273)
Description: Percentage of participants with seroresponse (based on the pre-booster baseline) for pseudovirus nAb ID50 against Omicron BA.1 Variant (B.1.1.529) at Days 181 and 366 are reported. Seroresponse was defined as a change from below the LLOQ to equal above 4 * LLOQ, or at least a 4-fold rise if baseline is equal to or above the LLOQ. LLOQ was 19.85 AU/mL and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529.
Time Frame: Days 181 and 366
Population: as for outcome 41
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Part G: mRNA-1273.214 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 308 | 239
percentage of participants
  Day 181 | 40.9 [35.4 to 46.6] | 25.9 [20.5 to 32.0]
  Day 366: number analyzed (Participants) | 193 | 179
  Day 366 | 52.8 [45.6 to 60.1] | 44.7 [37.3 to 52.3]
Statistical Analysis 1: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; SRR Difference = 14.5, 95% CI 2-sided [6.7 to 22.3] — Omicron BA.1 Variant (B.1.1.529) nAb at Day 181: Part G versus Part F (Cohort 2) mRNA-1273
Statistical Analysis 2: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; SRR Difference = 8.0, 95% CI 2-sided [-2.1 to 18.0] — Omicron BA.1 Variant (B.1.1.529) nAb at Day 366: Part G versus Part F (Cohort 2) mRNA-1273

43. Secondary Outcome: GMT of Serum Pseudovirus nAb ID50 Titers Against Omicron BA.1 Variant (B.1.1.529) and Ancestral SARS-CoV-2 (D614G) on Days 181 and 366 - mRNA-1273.214 (Part G) and mRNA-1273 (Part F, Cohort 2, 50 μg mRNA-1273)
Description: GMT of serum pseudovirus nAb ID50 titers against Omicron BA.1 Variant (B.1.1.529) and ancestral SARS-CoV-2 (D614G) on Days 181 and 366 is reported. Antibody values reported as below the LLOQ were replaced by 0.5 * LLOQ. Values greater than the ULOQ were replaced by the ULOQ if actual values were not available. LLOQ was 19.85 AU/mL and ULOQ was 15502.7 AU/mL for ID50 titer against B.1.1.529. LLOQ was 18.5 AU/mL and ULOQ was 45118 AU/mL for ID50 titer against ancestral SARS-CoV-2.
Time Frame: Days 181 and 366
Population: PPIS-Neg included all participants who received study injection; had pre-booster and Day 29 nAb data; had no major protocol deviations that impacted key or critical data; had no previous HIV infection; and who had no serologic or virologic evidence of SARS-CoV-2 infection at baseline. 'Overall number of participants analyzed' = participants evaluable for this outcome measure. 'Number analyzed' = participants evaluable for specified category.
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Part G: mRNA-1273.214 50 μg | Part F (Cohort 2): mRNA-1273 50 μg
Number analyzed (Participants) | 308 | 239
titer
  SARS-CoV-2 (B.1.1.529) nAb: Day 181 | 1044.9 [853.5 to 1279.2] | 693.7 [550.7 to 873.9]
  SARS-CoV-2 (D614G) nAb: Day 181 | 2683.2 [2300.6 to 3129.5] | 2393.3 [2047.4 to 2797.6]
  SARS-CoV-2 (B.1.1.529) nAb: Day 366: number analyzed (Participants) | 193 | 179
  SARS-CoV-2 (B.1.1.529) nAb: Day 366 | 1364.6 [1050.0 to 1773.6] | 1019.7 [776.3 to 1339.4]
  SARS-CoV-2 (D614G) nAb: Day 366: number analyzed (Participants) | 193 | 179
  SARS-CoV-2 (D614G) nAb: Day 366 | 2679.5 [2157.6 to 3327.5] | 2492.3 [2032.3 to 3056.5]
Statistical Analysis 1: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; GMR = 1.637, 95% CI 2-sided [1.243 to 2.155] — SARS-CoV-2 (B.1.1.529) nAb at Day 181: Part G versus Part F (Cohort 2) mRNA-1273
Statistical Analysis 2: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; GMR = 1.373, 95% CI 2-sided [0.953 to 1.976] — SARS-CoV-2 (B.1.1.529) nAb at Day 366: Part G versus Part F (Cohort 2) mRNA-1273
Statistical Analysis 3: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; GMR = 1.271, 95% CI 2-sided [1.051 to 1.537] — SARS-CoV-2 (D614G) nAb at Day 181: Part G versus Part F (Cohort 2) mRNA-1273
Statistical Analysis 4: Comparison: Part G: mRNA-1273.214 50 μg vs Part F (Cohort 2): mRNA-1273 50 μg; Test type: Other; GMR = 1.101, 95% CI 2-sided [0.830 to 1.461] — SARS-CoV-2 (D614G) nAb at Day 366: Part G versus Part F (Cohort 2) mRNA-1273

ADVERSE EVENTS:
Time Frame: Day 1 up to the end of the study (Day 366 for Parts A.1, B, C, D, F, and G; Day 181 for Parts A.2, H, J)
Description: The all-cause mortality was based on the full analysis set. The serious and other (not including serious) adverse events were based on the safety set which consisted of all participants who received the study vaccination.
Groups:
- Part A.1: mRNA-1273.211 50 µg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (COVE), received a single intramuscular (IM) booster dose of 50 micrograms (µg) of mRNA-1273.211 on Day 1 of Part A.1
- Part A.1: mRNA-1273.211 100 µg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (COVE), received a single IM booster dose of 100 µg of mRNA-1273.211 on Day 1 of Part A.1
- Part A.2: mRNA-1273.214 50 µg: Participants who had previously received 2 doses of mRNA-1273 as a primary series and a first booster dose of 50 µg of the mRNA-1273.211 in Part A.1 of this study, received a second IM booster dose of 50 µg of mRNA-1273.214 on Day 1 of Part A.2
- Part B: mRNA-1273 100 µg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (COVE), received a single IM booster dose of 100 µg of mRNA-1273 on Day 1 of Part B
- Part C: mRNA-1273.617.2 50 µg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (COVE) or under the EUA, received a single IM booster dose of 50 µg of mRNA-1273.617.2 on Day 1 of Part C
- Part C: mRNA-1273.617.2 100 µg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (COVE) or under the EUA, received a single IM booster dose of 100 µg of mRNA-1273.617.2 on Day 1 of Part C
- Part D: mRNA-1273.213 50 µg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (COVE) or under the EUA, received a single IM booster dose of 50 µg of mRNA-1273.213 on Day 1 of Part D
- Part D: mRNA-1273.213 100 µg: Participants who had previously received 2 doses of mRNA-1273 as a primary series in Study mRNA-1273-P301 (COVE) or under the EUA, received a single IM booster dose of 100 µg of mRNA-1273.213 on Day 1 of Part D
- Part E: mRNA-1273.213 100 µg: Participants who had previously received 2 doses of any SARS-CoV-2 mRNA authorized vaccine as a primary series (with a subset of enrolled participants who previously received Moderna's mRNA-1273 authorized vaccine as a primary series), received a single IM booster dose of 100 µg of mRNA-1273.213 on Day 1 of Part E
- Part F (Cohort 1): mRNA-1273.529 50 µg: Participants who had previously received 2 doses of mRNA-1273 as a primary series, received a single IM booster dose of 50 µg of mRNA-1273.529 on Day 1 of Part F
- Part F (Cohort 2): mRNA-1273 50 µg: Participants who had previously received 2 doses of mRNA-1273 100 µg as a primary series and a single booster dose of mRNA-1273 50 µg, received a second IM booster dose of 50 µg of mRNA-1273 on Day 1 of Part F
- Part F (Cohort 2): mRNA-1273.529 50 µg: Participants who had previously received 2 doses of mRNA-1273 100 µg as a primary series and a single booster dose of mRNA-1273 50 µg, received a second IM booster dose of 50 µg of mRNA-1273.529 on Day 1 of Part F
- Part G: mRNA-1273.214 50 µg: Participants who had previously received 2 doses of mRNA-1273 100 µg as a primary series and a single booster dose of mRNA-1273 50 µg, received a second IM booster dose of mRNA-1273.214 50 µg on Day 1 of Part G
- Part H: mRNA-1273.222 50 µg: Participants who had previously received 2 doses of mRNA-1273 100 µg as a primary series and a single booster dose of mRNA-1273 50 µg, received a second IM booster dose of 50 µg of mRNA-1273.222 on Day 1 of Part H
- Part J: mRNA-1273.231 50 µg: Participants who previously received a primary series of mRNA vaccine, a first booster dose of a monovalent mRNA vaccine, and a second booster dose of a bivalent mRNA vaccine against SARS-CoV-2, received a third IM booster dose of 50 µg of mRNA-1273.231 on Day 1 of Part J
- Part J: mRNA-1273.815 50 µg: Participants who previously received a primary series of mRNA vaccine, a first booster dose of a monovalent mRNA vaccine, and a second booster dose of a bivalent mRNA vaccine against SARS-CoV-2, received a third IM booster dose of 50 µg of mRNA-1273.815 on Day 1 of Part J
Arm/Group | Part A.1: mRNA-1273.211 50 µg | Part A.1: mRNA-1273.211 100 µg | Part A.2: mRNA-1273.214 50 µg | Part B: mRNA-1273 100 µg | Part C: mRNA-1273.617.2 50 µg | Part C: mRNA-1273.617.2 100 µg | Part D: mRNA-1273.213 50 µg | Part D: mRNA-1273.213 100 µg | Part E: mRNA-1273.213 100 µg | Part F (Cohort 1): mRNA-1273.529 50 µg | Part F (Cohort 2): mRNA-1273 50 µg | Part F (Cohort 2): mRNA-1273.529 50 µg | Part G: mRNA-1273.214 50 µg | Part H: mRNA-1273.222 50 µg | Part J: mRNA-1273.231 50 µg | Part J: mRNA-1273.815 50 µg
All-Cause Mortality (participants affected / at risk) | 1/300 | 0/593 | 0/135 | 1/305 | 0/581 | 1/586 | 0/327 | 0/583 | 0/42 | 0/133 | 2/376 | 0/375 | 2/437 | 2/510 | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 6/300 | 26/593 | 3/135 | 15/305 | 27/581 | 12/586 | 8/327 | 18/583 | 0/42 | 2/133 | 20/376 | 16/375 | 23/437 | 12/510 | 3/50 | 2/50
Other Adverse Events (participants affected / at risk) | 133/300 | 275/593 | 38/135 | 144/305 | 288/581 | 329/586 | 188/327 | 309/583 | 34/42 | 57/133 | 193/376 | 188/375 | 224/437 | 178/510 | 13/50 | 11/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A.1: mRNA-1273.211 50 µg (N=300) | Part A.1: mRNA-1273.211 100 µg (N=593) | Part A.2: mRNA-1273.214 50 µg (N=135) | Part B: mRNA-1273 100 µg (N=305) | Part C: mRNA-1273.617.2 50 µg (N=581) | Part C: mRNA-1273.617.2 100 µg (N=586) | Part D: mRNA-1273.213 50 µg (N=327) | Part D: mRNA-1273.213 100 µg (N=583) | Part E: mRNA-1273.213 100 µg (N=42) | Part F (Cohort 1): mRNA-1273.529 50 µg (N=133) | Part F (Cohort 2): mRNA-1273 50 µg (N=376) | Part F (Cohort 2): mRNA-1273.529 50 µg (N=375) | Part G: mRNA-1273.214 50 µg (N=437) | Part H: mRNA-1273.222 50 µg (N=510) | Part J: mRNA-1273.231 50 µg (N=50) | Part J: mRNA-1273.815 50 µg (N=50)
Abscess bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Campylobacter colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candida infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colonic abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Fungaemia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gangrene (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neurosyphilis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteomyelitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pelvic inflammatory disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia legionella (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rotavirus infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Septic shock (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tubo-ovarian abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urosepsis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemangioma of liver (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ovarian cancer stage IV (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleomorphic malignant fibrous histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Renal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alcohol abuse (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bipolar disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcoholic seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Amyotrophic lateral sclerosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aqueductal stenosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Facial paralysis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ischaemic cerebral infarction (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Migraine (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myelitis transverse (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paraesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal claudication (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vertigo positional (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute left ventricular failure (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Anginal equivalent (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 2 (3) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac disorder (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiogenic shock (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Coronary artery occlusion (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mitral valve incompetence (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocarditis (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accelerated hypertension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aortic stenosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Circulatory collapse (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haematoma (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertensive urgency (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Iliac artery occlusion (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pickwickian syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary artery thrombosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcoholic pancreatitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulum intestinal haemorrhagic (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematochezia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hiatus hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ileal stenosis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Incarcerated umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Intra-abdominal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mallory-Weiss syndrome (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Umbilical hernia, obstructive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Volvulus (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Alcoholic liver disease (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bile duct stone (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hepatic cyst (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angioedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Intervertebral disc degeneration (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sacroiliitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spinal synovial cyst (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Nephritis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Renal vascular thrombosis (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Adnexal torsion (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Menometrorrhagia (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Uterine prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Uterovaginal prolapse (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Non-cardiac chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Peripheral swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vascular stent thrombosis (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myocardial necrosis marker increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Staphylococcus test positive (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Transaminases increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Jaw fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint dislocation (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Wrist fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Device failure (Product Issues) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part A.1: mRNA-1273.211 50 µg (N=300) | Part A.1: mRNA-1273.211 100 µg (N=593) | Part A.2: mRNA-1273.214 50 µg (N=135) | Part B: mRNA-1273 100 µg (N=305) | Part C: mRNA-1273.617.2 50 µg (N=581) | Part C: mRNA-1273.617.2 100 µg (N=586) | Part D: mRNA-1273.213 50 µg (N=327) | Part D: mRNA-1273.213 100 µg (N=583) | Part E: mRNA-1273.213 100 µg (N=42) | Part F (Cohort 1): mRNA-1273.529 50 µg (N=133) | Part F (Cohort 2): mRNA-1273 50 µg (N=376) | Part F (Cohort 2): mRNA-1273.529 50 µg (N=375) | Part G: mRNA-1273.214 50 µg (N=437) | Part H: mRNA-1273.222 50 µg (N=510) | Part J: mRNA-1273.231 50 µg (N=50) | Part J: mRNA-1273.815 50 µg (N=50)
Asymptomatic COVID-19 (Infections and infestations) | 14 (15) | 40 (41) | 7 (7) | 20 (21) | 28 (28) | 21 (22) | 33 (34) | 14 (14) | 5 (5) | 12 (13) | 21 (21) | 27 (27) | 18 (19) | 24 (24) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 4 (4) | 6 (6) | 0 (0) | 16 (17) | 5 (5) | 7 (7) | 5 (5) | 24 (26) | 1 (1) | 2 (2) | 7 (7) | 5 (5) | 8 (8) | 4 (4) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 76 (76) | 143 (144) | 21 (21) | 87 (90) | 195 (201) | 227 (235) | 117 (124) | 220 (226) | 18 (18) | 30 (30) | 127 (132) | 119 (121) | 160 (164) | 74 (76) | 5 (5) | 2 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 16 (20) | 2 (2) | 8 (9) | 0 (0) | 4 (4) | 4 (4) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 6 (6) | 0 (0) | 0 (0)
Rhinovirus infection (Infections and infestations) | 14 (16) | 19 (20) | 4 (4) | 9 (10) | 22 (24) | 36 (39) | 11 (11) | 25 (26) | 3 (3) | 5 (5) | 18 (19) | 11 (12) | 27 (28) | 25 (27) | 3 (3) | 5 (6)
Upper respiratory tract infection (Infections and infestations) | 27 (28) | 63 (79) | 6 (6) | 21 (22) | 49 (62) | 49 (57) | 38 (51) | 53 (61) | 15 (15) | 9 (10) | 33 (41) | 31 (36) | 36 (39) | 36 (38) | 4 (4) | 2 (3)
Headache (Nervous system disorders) | 6 (7) | 24 (24) | 3 (3) | 6 (6) | 27 (30) | 32 (34) | 10 (11) | 24 (25) | 1 (1) | 12 (12) | 9 (13) | 15 (18) | 11 (11) | 21 (22) | 2 (2) | 1 (1)
Hypertension (Vascular disorders) | 12 (12) | 20 (22) | 0 (0) | 10 (12) | 13 (13) | 20 (20) | 17 (17) | 11 (12) | 0 (0) | 3 (3) | 18 (18) | 16 (16) | 13 (13) | 8 (8) | 1 (1) | 1 (1)
Respiratory disorder (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 4 (6) | 0 (0) | 0 (0) | 3 (3) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
Fatigue (General disorders) | 12 (14) | 36 (38) | 4 (4) | 6 (6) | 30 (34) | 29 (31) | 24 (25) | 33 (35) | 0 (0) | 11 (12) | 18 (20) | 17 (20) | 15 (17) | 25 (26) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2023-10-10): https://cdn.clinicaltrials.gov/large-docs/65/NCT04927065/Prot_000.pdf
  • Statistical Analysis Plan (2024-01-09): https://cdn.clinicaltrials.gov/large-docs/65/NCT04927065/SAP_001.pdf